CLINICAL TRIAL: NCT00348140
Title: A 54 Week, Double-blind, Randomised, Placebo-controlled, Parallel Group Study to Investigate the Effects of Rosiglitazone (Extended Release Tablets) as Adjunctive Therapy to Acetylcholinesterase Inhibitors on Cognition and Overall Clinical Response in APOE4-stratified Subjects With Mild to Moderate Alzheimer's Disease
Brief Title: Rosiglitazone (Extended Release Tablets) As Adjunctive Therapy In Subjects With Mild To Moderate Alzheimer's Disease
Acronym: REFLECT-3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AVA102670
Record Dates: First submitted 2006-06-30; First posted 2006-07-04 (Estimated); Results first posted 2017-09-05 (Actual); Last update posted 2017-09-05 (Actual); Status verified 2017-08

CONDITIONS: Alzheimer's Disease
Keywords: adjunctive therapy; moderate; Alzheimer's disease; apolipoprotein E; mild; rosiglitazone; cognition
MeSH Terms: conditions — Alzheimer Disease; Lymphoma, Follicular

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm 1 (Experimental): Rosiglitazone Extended Release 2mg OD
  Interventions: Drug: Rosiglitazone Extended Release 2mg
- Arm 2 (Experimental): Rosiglitazone Extended Release 8mg OD
  Interventions: Drug: Rosiglitazone Extended Release 8mg
- Arm 3 (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Rosiglitazone Extended Release 2mg — Rosiglitazone Extended Release 2mg OD
  Arms: Arm 1
Drug: Rosiglitazone Extended Release 8mg — Rosiglitazone Extended Release 8mg OD
  Arms: Arm 2
Other: Placebo — Placebo
  Arms: Arm 3

SUMMARY:
Rosiglitazone (RSG) has been tested in clinical studies and is approved by the FDA as a treatment for type II diabetes mellitus, a disease that occurs when the body is unable to effectively use glucose. RSG XR, the investigational drug used in this study, is an extended-release form of RSG.

This study tests whether RSG XR safely provides clinical benefit to people with mild to moderate Alzheimer's disease (AD) when combined with one of the currently approved AD medications, Aricept®, Razadyne® or Exelon®. RSG XR is a new approach to AD therapy and this study tests a new way to treat AD by testing whether one's genetic makeup affects the response to the study drug. Clinical data suggesting that RSG may benefit AD patients was first seen in a small study performed at the University of Washington and then from a larger GSK study conducted in Europe and New Zealand. In the first study, subjects receiving RSG once daily for 6 months scored significantly better on 3 tests of memory and thought than those who did not receive RSG. In the GSK study, those that appeared to benefit most from treatment with RSG XR had a specific genetic pattern. They did not have the gene that caused them to produce the protein apolipoprotein E e4 (APOE e4). Subjects who have the APOE e4 gene may have two copies, one from each parent, or they may have only one APOE e4 gene meaning that they inherited either the APOE e2 or APOE e3 version of the gene, instead of APOE e4, from one of their parents. Subjects with one copy of the APOE e4 gene remained at their same level of thinking ability while those with two copies of the APOE e4 gene, continued to worsen during the 6-month treatment. The current study will more directly test the effectiveness or RSG XR on people who either have or lack the APOE e4 gene.

DETAILED DESCRIPTION:
A 54-week, double-blind, randomized, placebo-controlled, parallel-group study to investigate the effects of rosiglitazone (extended release tablets) as adjunctive therapy to acetylcholinesterase inhibitors on cognition and overall clinical response in APOE e4-stratified subjects with mild to moderate Alzheimer's disease (REFLECT-3)

ELIGIBILITY:
Inclusion Criteria:

A subject will be eligible for inclusion in this study only if all of the following criteria apply:

* Male or female subject with a clinical diagnosis of probable Alzheimer's disease in accordance with NINCDS-ADRDA criteria (Appendix 2).

(Note: National Institute of Neurological and Communicative Disorders and Stroke (NINCDS) and Alzheimer's Disease and Related Disorders Association (ADRDA).)

* Subject has mild to moderate Alzheimer's disease as defined by a MMSE score 10 to 26 inclusive at Screening.
* Hachinski Ischemia Score ≤ 4 at Screening (See Appendix 3).
* Age ≥50 and ≤90 years.
* At least 6 months of ongoing acetylcholinesterase inhibitor therapy for Alzheimer's disease, with stable dosing for at least the last 2 months (and with no intent to change for the duration of the study).
* Current use of medication is in accordance with the criteria listed in Table 2 (Permitted Medications, Section 8.1).
* Female subjects must be post-menopausal (i.e. >1 year without menstrual period), surgically sterile, or agree to use adequate method of contraception (Appendix 4) for the duration of the study. Female subjects who are pre-menopausal or who have been post-menopausal for <1 year must undertake pregnancy testing (urine test) at Visit 1, which must be negative.
* Brain CT or MRI scan performed within the past 12 months or at Screening, showing no evidence of any other potential cause of dementia other than Alzheimer's disease.

(Note: Questionable CT or MRI scans should be discussed with the medical monitor, using central imaging guidelines.)

* Neurological exam without focal changes (excluding changes attributable to AD or peripheral trauma).
* Subject has the ability to comply with procedures for cognitive and other testing.
* Subject lives with (or has substantial periods of contact with) a regular caregiver who is willing to attend all visits, oversee the subject's compliance with protocol-specified procedures and study medication, and report on subject's status.

(Note: A non-cohabiting caregiver must spend sufficient time with the subject so that, in the opinion of the Investigator, the caregiver can reliably assess cognitive function, activities and behavior, and report on the subject's compliance and health. As caregiver time spent with a potential subject is anticipated to be highly variable across countries and cultures, GSK will consider a variety of different measures by which this stipulation may be met, and GSK should be consulted if adequacy of a caregiver situation is in doubt. However, as guidance, the ability for a caregiver to meet his/her expected responsibilities for this study would normally be possible when the caregiver spends no less than 10 hours per week with the subject, divided over multiple days.)

* Subject has provided full written informed consent prior to the performance of any protocol-specified procedure; or if unable to provide informed consent due to cognitive status, full written informed consent on behalf of the subject has been provided by a legally acceptable representative.

(Note: Consent by legally acceptable representative is allowed where this is in accordance with local laws, regulations and ethics committee policy.)

* Caregiver has provided full written informed consent on his/her own behalf prior to the performance of any protocol-specified procedure.
* Subjects considered for enrolment must have a QTc (either QTc B (Bazett's correction) or QTc F (Fridericia's correction)) <450msec at Visit 1, with the exception of subjects with bundle branch block (for whom either QTc B or QTc F must be <480msec).

(Note: For the purposes of these criteria, QTc B is defined as (QT interval [msec]) / (square root of RR interval [seconds]); and QTc F is defined as (QT interval [msec]) / (cube root of RR interval [seconds]).)

Exclusion Criteria:

A subject will not be eligible for inclusion in this study if any of the following criteria apply:

* Diagnosis of possible, probable, or definite vascular dementia in accordance with NINDS-AIREN criteria (Appendix 5).

(Note: National Institute of Neurological Disorders and Stroke (NINDS) and Association Internationale pour la Recherche et l'Enseignement en Neurosciences (AIREN).)

* History or evidence of any other CNS disorder that could be interpreted as a cause of dementia: e.g. cerebrovascular disease (stroke, hemorrhage), structural abnormality, epilepsy, infectious or inflammatory/demyelinating CNS conditions, Parkinson's disease.
* Evidence of the following disorders: current vitamin B12 deficiency, positive syphilis serology, or active thyroid dysfunction (particularly that suggestive of hypothyroidism), including abnormally high or low serum levels of thyroid stimulating hormone (TSH), that are clinically significant in the opinion of the investigator.

(Note: Testing is required for each parameter only when no result is available from previous 12 months.)

* History of Type 1 diabetes mellitus or secondary diabetes mellitus.
* Type 2 diabetes mellitus where the subject is being treated with insulin, a PPARγ agonist, or an insulin secretagogue (e.g. a sulfonylurea or glitinide).
* Any patient with an HbA1c ≥8.5%. (See Section 6.3.8.4 for Safety Measures for Enrolled Subjects with Type 2 Diabetes Mellitus.)
* History or clinical/investigational evidence of congestive heart failure defined by the New York Heart Association criteria (Class I to IV cardiac status; Appendix 6).
* History of cardiovascular event within the last 6 months (i.e. intervention, percutaneous coronary intervention, vascular surgery, acute coronary syndrome [non Q-wave myocardial infarction, Q-wave myocardial infarction, unstable angina] or significant arrhythmia; or major intervention (e.g. cardiac surgery or angiography plus stenting) scheduled).
* History of significant psychiatric illness such as schizophrenia or bipolar affective disorder that in the opinion of the Investigator would interfere with participation in the study, major depressive disorder (according to DSM-IV) in the past year, or current active depression requiring initiation of treatment.

(Note: If not currently treated, but active depression is suspected, the Cornell Scale for Depression in Dementia (CSDD, Appendix 7) can be used by the Investigator as a guide for deciding whether a prospective subject requires treatment. If the subject has a CSDD score >7, the Investigator should decide if the subject has depression in need of prescribed medication, and a CSDD >12 is considered a strong indicator that treatment is needed. Subjects will be allowed to re-screen after their depression has been adequately managed for >3 months.)

* History or presence of gastro-intestinal, hepatic, or renal disease or other condition known to interfere with the absorption, distribution, metabolism, or excretion of drugs, or any other clinically relevant abnormality, medical or psychiatric condition, which, in the opinion of the Investigator, makes the subject unsuitable for inclusion in the study.
* Clinically significant peripheral edema at the time of screening.
* Current or recent drug or alcohol abuse or dependence (defined by DSM-IV criteria for substance-related disorders), or recent or remote history of the same if that could be a contributing factor to the dementia.
* Systolic blood pressure >165 or <90 mmHg or diastolic blood pressure >95 or <60 mmHg at the time of screening.
* Clinically significant anemia (i.e. hemoglobin <11 g/dL for males or <10 g/dL for females) or presence of hemoglobinopathies which would prevent accurate assessment of HbA1c.
* Abnormal kidney function tests (>1.5 times the upper limit of normal (ULN)).
* ALT, AST, or alkaline phosphatase values >2.5 times the ULN, total bilirubin values >1.5 times the ULN, or history of severe hepatobiliary disease (e.g. hepatitis B or C, or cirrhosis, Child-Pugh Class B/C).

(Note: For subjects with a diagnosis of Gilberts Syndrome and an isolated increase in total bilirubin >1.5 ULN, fractionation should be performed. If all of the following conditions are met, the patient may enter or remain in the study, even if total bilirubin >1.5 ULN:

* an elevated unconjugated (indirect) bilirubin;
* the percentage of direct bilirubin <35%;
* ALT, AST, and alkaline phosphatase <2.5 ULN if subject is in screening (<2.0 ULN for Canadian subjects only), or ≤3 ULN if subject is already randomized into the study)
* History of a bone marrow transplant.
* Subject is unable (with assistance, if appropriate) to take study medication as prescribed throughout the study or is at risk of non-compliance with study medication or procedures.
* Subject is an immediate family member or employee of the participating Investigator, of any of the participating site staff, or of GSK.
* In France, a subject is neither affiliated with nor a beneficiary of a social security category.
* The French subject has participated in any study using an investigational drug during the previous 30 days or 5 half-lives (whichever is longer).
* Cognitive tasks prescribed for cognitive rehabilitation and performed under medical supervision are prohibited for 6 months prior to Screening, as well as for the duration of the study.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1468 (Actual)
Dates: Start 2006-07-12 (Actual); Primary Completion 2009-03-20 (Actual); Study Completion 2009-03-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (161):
- United States (47):
  - GSK Investigational Site, Sun City, Arizona
  - GSK Investigational Site, Tucson, Arizona
  - GSK Investigational Site, Little Rock, Arkansas
  - GSK Investigational Site, Laguna Hills, California
  - GSK Investigational Site, Redlands, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, San Francisco, California
  - GSK Investigational Site, Norwalk, Connecticut
  - GSK Investigational Site, Deerfield Beach, Florida
  - GSK Investigational Site, Delray Beach, Florida
  - GSK Investigational Site, Fort Lauderdale, Florida
  - GSK Investigational Site, Hialeah, Florida
  - GSK Investigational Site, Ocala, Florida
  - GSK Investigational Site, St. Petersburg, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, Decatur, Georgia
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Springfield, Massachusetts
  - GSK Investigational Site, West Yarmouth, Massachusetts
  - GSK Investigational Site, Eatontown, New Jersey
  - GSK Investigational Site, Toms River, New Jersey
  - GSK Investigational Site, Whiting, New Jersey
  - GSK Investigational Site, Amherst, New York
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Rochester, New York
  - GSK Investigational Site, Syracuse, New York
  - GSK Investigational Site, Raleigh, North Carolina
  - GSK Investigational Site, Winston-Salem, North Carolina
  - GSK Investigational Site, Centerville, Ohio
  - GSK Investigational Site, Columbus, Ohio
  - GSK Investigational Site, Toledo, Ohio
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Tulsa, Oklahoma
  - GSK Investigational Site, Jenkintown, Pennsylvania
  - GSK Investigational Site, Norristown, Pennsylvania
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, East Providence, Rhode Island
  - GSK Investigational Site, Providence, Rhode Island
  - GSK Investigational Site, Greer, South Carolina
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Wichita Falls, Texas
  - GSK Investigational Site, Salt Lake City, Utah
  - GSK Investigational Site, Charlottesville, Virginia
  - GSK Investigational Site, Seattle, Washington
  - GSK Investigational Site, Middleton, Wisconsin
  - GSK Investigational Site, Milwaukee, Wisconsin
- Australia (11):
  - GSK Investigational Site, Hornsby, New South Wales
  - GSK Investigational Site, Randwick, New South Wales
  - GSK Investigational Site, Auchenflower, Queensland
  - GSK Investigational Site, Chermside, Queensland
  - GSK Investigational Site, Kippa-Ring, Queensland
  - GSK Investigational Site, Adelaide, South Australia
  - GSK Investigational Site, Woodville, South Australia
  - GSK Investigational Site, Cheltenham, Victoria
  - GSK Investigational Site, Heidelberg West, Victoria
  - GSK Investigational Site, Kew, Victoria
  - GSK Investigational Site, Nedlands, Western Australia
- Belgium (4):
  - GSK Investigational Site, Brussels
  - GSK Investigational Site, Kortrijk
  - GSK Investigational Site, Leuven
  - GSK Investigational Site, Woluwe-Saint-Lambert
- Bulgaria (2):
  - GSK Investigational Site, Sofia
  - GSK Investigational Site, Varna
- Canada (12):
  - GSK Investigational Site, Kelowna, British Columbia
  - GSK Investigational Site, Saint John, New Brunswick
  - GSK Investigational Site, Kentville, Nova Scotia
  - GSK Investigational Site, Kingston, Ontario
  - GSK Investigational Site, Ottawa, Ontario
  - GSK Investigational Site, Peterborough, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Greenfield Park, Quebec
  - GSK Investigational Site, Mirabel, Quebec
  - GSK Investigational Site, Montreal, Quebec
  - GSK Investigational Site, Sherbrooke, Quebec
  - GSK Investigational Site, Québec
- Czechia (3):
  - GSK Investigational Site, Olomouc
  - GSK Investigational Site, Prague
  - GSK Investigational Site, Trutnov
- Finland (3):
  - GSK Investigational Site, Helsinki
  - GSK Investigational Site, Joensuu
  - GSK Investigational Site, Kuopio
- France (12):
  - GSK Investigational Site, Bordeaux
  - GSK Investigational Site, La Chapelle-sur-Erdre
  - GSK Investigational Site, La Seyne-sur-Mer
  - GSK Investigational Site, Lille
  - GSK Investigational Site, Limoges
  - GSK Investigational Site, Metz
  - GSK Investigational Site, Nantes
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Sautron
  - GSK Investigational Site, Toulon
  - GSK Investigational Site, Toulouse
  - GSK Investigational Site, Valence
- Germany (20):
  - GSK Investigational Site, Aalen, Baden-Wurttemberg
  - GSK Investigational Site, Calw, Baden-Wurttemberg
  - GSK Investigational Site, Ellwangen, Baden-Wurttemberg
  - GSK Investigational Site, Ludwigsburg, Baden-Wurttemberg
  - GSK Investigational Site, Stuttgart, Baden-Wurttemberg
  - GSK Investigational Site, Tübingen, Baden-Wurttemberg
  - GSK Investigational Site, Ulm, Baden-Wurttemberg
  - GSK Investigational Site, Wiesloch, Baden-Wurttemberg
  - GSK Investigational Site, Alzenau in Unterfranken, Bavaria
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Unterhaching, Bavaria
  - GSK Investigational Site, Bad Saarow, Brandenburg
  - GSK Investigational Site, Bad Homburg, Hesse
  - GSK Investigational Site, Erbach im Odenwald, Hesse
  - GSK Investigational Site, Chemnitz, Saxony
  - GSK Investigational Site, Dresden, Saxony
  - GSK Investigational Site, Leipzig, Saxony
  - GSK Investigational Site, Gera, Thuringia
  - GSK Investigational Site, Jena, Thuringia
  - GSK Investigational Site, Berlin
- Hong Kong (2):
  - GSK Investigational Site, Hong Kong
  - GSK Investigational Site, Shatin
- Malaysia (3):
  - GSK Investigational Site, Bandar Tun Razak, Cheras
  - GSK Investigational Site, Ipoh
  - GSK Investigational Site, Kelantan
- Netherlands (6):
  - GSK Investigational Site, 's-Hertogenbosch
  - GSK Investigational Site, Alkmaar
  - GSK Investigational Site, Blaricum
  - GSK Investigational Site, Hengelo
  - GSK Investigational Site, Hilversum
  - GSK Investigational Site, The Hague
- Philippines (2):
  - GSK Investigational Site, Manila
  - GSK Investigational Site, Pasig
- Poland (4):
  - GSK Investigational Site, Bydgoszcz
  - GSK Investigational Site, Krakow
  - GSK Investigational Site, Torun
  - GSK Investigational Site, Warsaw
- GSK Investigational Site, Singapore, Singapore
- Slovakia (2):
  - GSK Investigational Site, Bratislava
  - GSK Investigational Site, Košice
- Slovenia (2):
  - GSK Investigational Site, Ljubljana
  - GSK Investigational Site, Šempeter v Savinj. Dolini
- South Africa (7):
  - GSK Investigational Site, Loeventstein
  - GSK Investigational Site, Oakdale
  - GSK Investigational Site, Richards Bay
  - GSK Investigational Site, Rosebank
  - GSK Investigational Site, Somerset West
  - GSK Investigational Site, Waverley, Bloemfontein
  - GSK Investigational Site, Willows, X14, Pretoria
- South Korea (2):
  - GSK Investigational Site, Seongnam-si
  - GSK Investigational Site, Seoul
- Spain (4):
  - GSK Investigational Site, Baracaldo/Vizcaya
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Palma de Mallorca
  - GSK Investigational Site, Tarrasa, Barcelona
- Sweden (6):
  - GSK Investigational Site, Falköping
  - GSK Investigational Site, Jönköping
  - GSK Investigational Site, Kalix
  - GSK Investigational Site, Mölndal
  - GSK Investigational Site, Sundsvall
  - GSK Investigational Site, Umeå
- United Kingdom (6):
  - GSK Investigational Site, Blackpool, Lancashire
  - GSK Investigational Site, Bradford
  - GSK Investigational Site, Liverpool
  - GSK Investigational Site, Stirling
  - GSK Investigational Site, West End, Southampton
  - GSK Investigational Site, West of Scotland Science Park, Glasgow

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Harrington C, Sawchak S, Chiang C, Davies J, Donovan C, Saunders AM, Irizarry M, Jeter B, Zvartau-Hind M, van Dyck CH, Gold M. Rosiglitazone does not improve cognition or global function when used as adjunctive therapy to AChE inhibitors in mild-to-moderate Alzheimer's disease: two phase 3 studies. Curr Alzheimer Res. 2011 Aug;8(5):592-606. doi: 10.2174/156720511796391935. PMID 21592048
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: AVA102670 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: AVA102670 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: AVA102670 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: AVA102670 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: AVA102670 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: AVA102670 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: AVA102670 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 1485 participants with Alzheimer's disease (AD) who were being treated with an approved Acetylcholinesterase inhibitor (AChEI) were randomized in the study and stratified by Apolipoprotein E gene (APOE) ε4 allele status. Total of 1468 were included in safety population and 1429 in the intent-to-treat population (ITT).
Groups:
- Placebo: Participants randomized to this arm received matching Rosiglitazone extended release (RSG XR) placebo tablets once daily which remained constant throughout the 48 Week treatment period. From Week 48 all the participants received single-blind placebo treatment as one tablet daily until Visit 10 (Week 54)
- RSG XR 2mg: Participants randomized to this arm received RSG XR 2 milligrams (mg) once daily which remained constant throughout the 48 Week treatment period. From Week 48 all the participants received single-blind placebo treatment as one tablet daily until Visit 10 (Week 54)
- RSG XR 8mg: Participants randomized to this arm received RSG XR 8 mg one 4mg tablet once daily for the first 4 weeks of treatment. From Visit 3 (Week 4) onwards, these participants received one 8mg tablet once daily for the remaining 44 weeks of double-blind treatment. From Week 48 all participants received single-blind placebo treatment as one tablet daily, until Visit 10 (Week 54)
Period: Overall Study
Arm/Group | Placebo | RSG XR 2mg | RSG XR 8mg
Started | 487 | 490 | 491
Completed | 361 | 351 | 328
Not Completed | 126 | 139 | 163
Not completed — Adverse Event | 46 | 49 | 78
Not completed — Lost to Follow-up | 4 | 4 | 4
Not completed — Protocol Violation | 12 | 13 | 14
Not completed — Withdrawal by Subject | 32 | 40 | 40
Not completed — Non-compliance | 8 | 13 | 5
Not completed — Participant at risk due to study drug | 2 | 0 | 0
Not completed — Conditional medication increased dose | 1 | 0 | 0
Not completed — Caregiver related | 4 | 7 | 3
Not completed — Participant hospitalised | 3 | 0 | 0
Not completed — Efficacy related | 1 | 1 | 0
Not completed — Administration related | 3 | 1 | 1
Not completed — Unmet inclusion-exclusion criteria | 1 | 0 | 1
Not completed — Participant unwell | 1 | 0 | 0
Not completed — Screen failure | 1 | 0 | 0
Not completed — Investigator decided to discontinue | 4 | 1 | 4
Not completed — Decided to discontinue on their own | 1 | 4 | 1
Not completed — Use of prohibited drug | 1 | 0 | 2
Not completed — Disease progression | 1 | 2 | 5
Not completed — Increased risk of cardiac infarction | 0 | 1 | 0
Not completed — Serious adverse event | 0 | 1 | 0
Not completed — Abnormal ECG | 0 | 1 | 3
Not completed — Participant died | 0 | 1 | 0
Not completed — Exclusion criteria met | 0 | 0 | 1
Not completed — Memory declined | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Participants randomized to this arm received matching RSG XR placebo tablets once daily which remained constant throughout the 48 Week treatment period. From Week 48 all the participants received single-blind placebo treatment as one tablet daily until Visit 10 (Week 54)
- RSG XR 2mg: Participants randomized to this arm received RSG XR 2 mg once daily which remained constant throughout the 48 Week treatment period. From Week 48 all the participants received single-blind placebo treatment as one tablet daily until Visit 10 (Week 54)
- Total: Total of all reporting groups
Arm/Group | Placebo | RSG XR 2mg | RSG XR 8mg | Total
Number analyzed (Participants) | 487 | 490 | 491 | 1468
Age, Continuous [Mean (Standard Deviation); unit: Years] | 72.8 (8.19) | 73.4 (8.19) | 73.6 (8.40) | 73.3 (8.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 272 | 276 | 268 | 816
  Male | 215 | 214 | 223 | 652
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 16 | 14 | 18 | 48
  Not Hispanic or Latino | 467 | 473 | 470 | 1410
  Missing | 4 | 3 | 3 | 10

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Alzheimer's Disease Assessment Scale - Cognitive Subscale (ADAS-Cog) Total Score at Week 48, as a Function of APOE ε4 Status in APOE4 Negatives Cohort
Description: The 11-item ADAS-Cog assessed a range of cognitive abilities including memory, comprehension, orientation in time and place and spontaneous speech. Most items were evaluated by tests, but some were dependent on clinician ratings on a five point scale. Scores range from 0 to 70 with higher scores indicating greater dysfunction. Change from Baseline was calculated as value at scheduled time point minus Baseline value. Baseline was defined as value at Week 0. Estimated value was calculated by Active treatment minus Placebo. The adjusted means were presented. A hierarchical testing procedure was used to control for statistical tests in the two RSG dose groups and the genetic subgroups.
Time Frame: Baseline (Week 0) and Week 48
Population: ITT population comprised of all participants randomized to treatment, who had taken at least one dose of study medication and who had at least one post baseline efficacy assessment. Number of participants with observed data contributing to the analysis have been presented.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | RSG XR 2mg | RSG XR 8mg
Number analyzed (Participants) | 145 | 142 | 137
Scores on a scale | 3.2 (0.54) | 3.5 (0.53) | 4.0 (0.63)
Statistical Analysis 1: Comparison: Placebo vs RSG XR 2mg; Test type: Superiority; p = 0.739, Mixed model for repeated measures; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Net) = 0.3, 95% CI 2-sided [-1.2 to 1.8] — Difference in adjusted least square means was shown (Active treatment minus Placebo); n = Number of participants with evaluable data
Statistical Analysis 2: Comparison: Placebo vs RSG XR 8mg; Test type: Superiority; p = 0.343, Mixed model for repeated measures; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Net) = 0.8, 95% CI 2-sided [-0.8 to 2.4] — [estimate comment as in outcome 1, analysis 1]

2. Primary Outcome: Change From Baseline in ADAS-Cog Total Score at Week 48, as a Function of APOE ε4 Status in All Except E4/E4s Cohort
Description: The 11-item ADAS-Cog assessed a range of cognitive abilities including memory, comprehension, orientation in time and place and spontaneous speech. Most items were evaluated by tests, but some were dependent on clinician ratings on a five point scale. Scores range from 0 to 70 with higher scores indicating greater dysfunction. Change from Baseline was calculated as value at scheduled time point minus Baseline value. Baseline was defined as value a t Week 0. Estimated value was calculated by Active treatment minus Placebo. The adjusted means were presented. A hierarchical testing procedure was used to control for statistical tests in the two RSG dose groups and the genetic subgroups.
Time Frame: Baseline (Week 0) and Week 48
Population: ITT population. Number of participants with observed data contributing to the analysis have been presented.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | RSG XR 2mg | RSG XR 8mg
Number analyzed (Participants) | 303 | 302 | 274
Scores on a scale | 3.8 (0.38) | 3.6 (0.35) | 3.8 (0.41)
Statistical Analysis 1: Comparison: Placebo vs RSG XR 2mg; Test type: Superiority; p = 0.783, Mixed model for repeated measures; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Net) = -0.1, 95% CI 2-sided [-1.1 to 0.9] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs RSG XR 8mg; Test type: Superiority; p = 0.940, Mixed model for repeated measures; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Net) = 0.0, 95% CI 2-sided [-1.1 to 1.1] — [estimate comment as in outcome 1, analysis 1]

3. Primary Outcome: Change From Baseline in ADAS-Cog Total Score at Week 48, as a Function of APOE ε4 Status in Full Population Cohort
Description: as for outcome 2
Time Frame: Baseline (Week 0) and Week 48
Population: ITT population. Number of participants with observed data contributing to the analysis have been presented.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | RSG XR 2mg | RSG XR 8mg
Number analyzed (Participants) | 361 | 343 | 331
Scores on a scale | 3.9 (0.35) | 3.8 (0.33) | 3.8 (0.36)
Statistical Analysis 1: Comparison: Placebo vs RSG XR 2mg; Test type: Superiority; p = 0.763, Mixed model for repeated measures; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Net) = -0.1, 95% CI 2-sided [-1.1 to 0.8] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs RSG XR 8mg; Test type: Superiority; p = 0.800, Mixed model for repeated measures; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Net) = -0.1, 95% CI 2-sided [-1.1 to 0.9] — [estimate comment as in outcome 1, analysis 1]

4. Primary Outcome: Change From Baseline in Clinical Dementia Rating Scale - Sum of Boxes (CDR-SB) Score at Week 48, as a Function of APOE ε4 Status in APOE4 Negatives Cohort
Description: The CDR-SB was a validated clinical assessment of global function in patients with AD. Impairment was scored in each of 6 cognitive categories on a scale in which none = 0, questionable = 0.5, mild = 1, moderate = 2, and severe = 3. The 6 individual category ratings, or "box scores", can be added together to give the CDR-Sum of Boxes which ranges from 0 to 18 (severe impairment). Change from Baseline was calculated as value at scheduled time point minus Baseline value. Baseline was defined as value a t Week 0. Estimated value was calculated by Active treatment minus Placebo. The adjusted means were presented. Primary inference will be based on the week 48 treatment differences obtained from the MMRM model. A hierarchical testing procedure was used to control for statistical tests in the two RSG dose groups and the genetic subgroups.
Time Frame: Baseline (Week 0) and Week 48
Population: ITT population. Number of participants with observed data contributing to the analysis have been presented.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | RSG XR 2mg | RSG XR 8mg
Number analyzed (Participants) | 146 | 144 | 138
Scores on a scale | 1.8 (0.20) | 1.7 (0.20) | 1.7 (0.17)
Statistical Analysis 1: Comparison: Placebo vs RSG XR 2mg; Test type: Superiority; p = 0.611, Mixed model for repeated measures; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Net) = -0.1, 95% CI 2-sided [-0.7 to 0.4] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs RSG XR 8mg; Test type: Superiority; p = 0.741, Mixed model for repeated measures; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Net) = -0.1, 95% CI 2-sided [-0.6 to 0.4] — [estimate comment as in outcome 1, analysis 1]

5. Primary Outcome: Change From Baseline in CDR-SB Score at Week 48, as a Function of APOE ε4 Status in All Except E4/E4s Cohort
Description: as for outcome 4
Time Frame: Baseline (Week 0) and Week 48
Population: ITT population. Number of participants with observed data contributing to the analysis have been presented.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | RSG XR 2mg | RSG XR 8mg
Number analyzed (Participants) | 302 | 311 | 272
Scores on a scale | 1.8 (0.13) | 1.8 (0.13) | 1.7 (0.13)
Statistical Analysis 1: Comparison: Placebo vs RSG XR 2mg; Test type: Superiority; p = 0.913, Mixed model for repeated measures; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Net) = 0.0, 95% CI 2-sided [-0.4 to 0.3] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs RSG XR 8mg; Test type: Superiority; p = 0.481, Mixed model for repeated measures; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Net) = -0.1, 95% CI 2-sided [-0.5 to 0.2] — [estimate comment as in outcome 1, analysis 1]

6. Primary Outcome: Change From Baseline in CDR-SB Score at Week 48, as a Function of APOE ε4 Status in Full Population Cohort
Description: as for outcome 4
Time Frame: Baseline (Week 0) and Week 48
Population: ITT population. Number of participants with observed data contributing to the analysis have been presented.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | RSG XR 2mg | RSG XR 8mg
Number analyzed (Participants) | 360 | 349 | 331
Scores on a scale | 1.9 (0.12) | 1.8 (0.13) | 1.8 (0.12)
Statistical Analysis 1: Comparison: Placebo vs RSG XR 2mg; Test type: Superiority; p = 0.557, Mixed model for repeated measures; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Net) = -0.1, 95% CI 2-sided [-0.4 to 0.2] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs RSG XR 8mg; Test type: Superiority; p = 0.404, Mixed model for repeated measures; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Net) = -0.1, 95% CI 2-sided [-0.5 to 0.2] — [estimate comment as in outcome 1, analysis 1]

7. Secondary Outcome: Change From Baseline in ADAS-Cog Total Score at Weeks 8, 16, 24 and 36
Description: The 11-item ADAS-Cog assessed a range of cognitive abilities including memory, comprehension, orientation in time and place and spontaneous speech. Most items were evaluated by tests, but some were dependent on clinician ratings on a five point scale. Scores range from 0 to 70 with higher scores indicating greater dysfunction. Change from Baseline was calculated as value at scheduled time point minus Baseline value. Baseline was defined as value a t Week 0. It was calculated at Weeks 8, 16, 24 and 36. Full population data was presented.
Time Frame: Baseline (Week 0) and Week 8, 16, 24, 36
Population: ITT population. Number of participants with observed data contributing to the analysis.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | RSG XR 2mg | RSG XR 8mg
Number analyzed (Participants) | 479 | 480 | 470
Scores on a scale
  Week 8: number analyzed (Participants) | 460 | 451 | 440
  Week 8 | 0.1 (0.23) | 0.2 (0.23) | 0.3 (0.23)
  Week 16: number analyzed (Participants) | 440 | 430 | 411
  Week 16 | 0.2 (0.24) | 0.3 (0.23) | 0.2 (0.24)
  Week 24: number analyzed (Participants) | 422 | 408 | 379
  Week 24 | 1.1 (0.26) | 1.5 (0.28) | 1.1 (0.27)
  Week 36: number analyzed (Participants) | 383 | 381 | 352
  Week 36 | 2.6 (0.31) | 2.8 (0.29) | 2.6 (0.31)
Statistical Analysis 1: Comparison: Placebo vs RSG XR 2mg; For Week 8; Test type: Superiority; p = 0.633, Mixed model for repeated measures; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Net) = 0.1, 95% CI 2-sided [-0.5 to 0.8] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs RSG XR 8mg; For Week 8; Test type: Superiority; p = 0.575, Mixed model for repeated measures; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Net) = 0.2, 95% CI 2-sided [-0.4 to 0.8] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs RSG XR 2mg; For Week 16; Test type: Superiority; p = 0.820, Mixed model for repeated measures; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Net) = 0.1, 95% CI 2-sided [-0.6 to 0.7] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Placebo vs RSG XR 8mg; For Week 16; Test type: Superiority; p = 0.908, Mixed model for repeated measures; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Net) = 0.0, 95% CI 2-sided [-0.7 to 0.6] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Placebo vs RSG XR 2mg; For Week 24; Test type: Superiority; p = 0.292, Mixed model for repeated measures; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Net) = 0.4, 95% CI 2-sided [-0.3 to 1.1] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Placebo vs RSG XR 8mg; For Week 24; Test type: Superiority; p = 0.978, Mixed model for repeated measures; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Net) = 0.0, 95% CI 2-sided [-0.7 to 0.7] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: Placebo vs RSG XR 2mg; For Week 36; Test type: Superiority; p = 0.691, Mixed model for repeated measures; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Net) = 0.2, 95% CI 2-sided [-0.6 to 1.0] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 8: Comparison: Placebo vs RSG XR 8mg; For Week 36; Test type: Superiority; p = 0.849, Mixed model for repeated measures; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Net) = -0.1, 95% CI 2-sided [-0.9 to 0.8] — [estimate comment as in outcome 1, analysis 1]

8. Secondary Outcome: Change From Baseline in CDR-SB Score at Weeks 12, 24 and 36
Description: The CDR-SB was a validated clinical assessment of global function in patients with AD. Impairment was scored in each of 6 cognitive categories on a scale in which none = 0, questionable = 0.5, mild = 1, moderate = 2, and severe = 3. The 6 individual category ratings, or "box scores", can be added together to give the CDR-Sum of Boxes which ranges from 0 to 18 (severe impairment). Change from Baseline was calculated as value at scheduled time point minus Baseline value. Baseline was defined as value a t Week 0. Estimated value was calculated by Active treatment minus Placebo. The adjusted means were presented. It was calculated at Weeks 12, 24 and 36. Full population data was presented.
Time Frame: Baseline (Week 0) and Week 12, 24, 36
Population: ITT population. Number of participants with observed data contributing to the analysis.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | RSG XR 2mg | RSG XR 8mg
Number analyzed (Participants) | 479 | 480 | 470
Scores on a scale
  Week 12: number analyzed (Participants) | 437 | 432 | 422
  Week 12 | 0.3 (0.07) | 0.4 (0.08) | 0.3 (0.07)
  Week 24: number analyzed (Participants) | 413 | 400 | 376
  Week 24 | 0.9 (0.10) | 0.8 (0.10) | 0.9 (0.09)
  Week 36: number analyzed (Participants) | 382 | 374 | 350
  Week 36 | 1.4 (0.11) | 1.3 (0.11) | 1.3 (0.10)
Statistical Analysis 1: Comparison: Placebo vs RSG XR 2mg; For Week 12; Test type: Superiority; p = 0.938, Mixed model for repeated measures; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Net) = 0.0, 95% CI 2-sided [-0.2 to 0.2] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs RSG XR 8mg; For Week 12; Test type: Superiority; p = 0.887, Mixed model for repeated measures; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Net) = 0.0, 95% CI 2-sided [-0.2 to 0.2] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs RSG XR 2mg; For Week 24; Test type: Superiority; p = 0.465, Mixed model for repeated measures; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Net) = -0.1, 95% CI 2-sided [-0.4 to 0.2] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Placebo vs RSG XR 8mg; For Week 24; Test type: Superiority; p = 0.596, Mixed model for repeated measures; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Net) = 0.1, 95% CI 2-sided [-0.2 to 0.3] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Placebo vs RSG XR 2mg; For Week 36; Test type: Superiority; p = 0.452, Mixed model for repeated measures; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Net) = -0.1, 95% CI 2-sided [-0.4 to 0.2] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Placebo vs RSG XR 8mg; For Week 36; Test type: Superiority; p = 0.429, Mixed model for repeated measures; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Net) = -0.1, 95% CI 2-sided [-0.4 to 0.2] — [estimate comment as in outcome 1, analysis 1]

9. Secondary Outcome: Change From Screening in Mini Mental State Examination (MMSE) Total Score
Description: The MMSE consists of 11 tests of orientation, memory (recent and immediate), concentration, language and praxis. Scores range from 0 to 30, with lower scores indicating greater cognitive impairment. The scale is completed by the investigator, based on the performance of the participant. Change from screening was calculated as value at scheduled time point minus screening value. Baseline was defined as value a t Week 0. Estimated value was calculated by Active treatment minus Placebo. The adjusted means were presented. Full population data was presented.
Time Frame: Screening (Week -4) and Week 48
Population: ITT population. Only those participants available at that particular time point were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | RSG XR 2mg | RSG XR 8mg
Number analyzed (Participants) | 366 | 356 | 336
Scores on a scale | -2.0 (0.21) | -2.3 (0.22) | -2.0 (0.22)
Statistical Analysis 1: Comparison: Placebo vs RSG XR 2mg; Test type: Superiority; p = 0.386, ANCOVA; Mean Difference (Net) = -0.3, 95% CI 2-sided [-0.8 to 0.3]
Statistical Analysis 2: Comparison: Placebo vs RSG XR 8mg; Test type: Superiority; p = 0.999, ANCOVA; Mean Difference (Net) = 0.0, 95% CI 2-sided [-0.6 to 0.6]

10. Secondary Outcome: Change From Baseline in Disability Assessment for Dementia (DAD) Total Score
Description: The DAD assessed the ability of a participant to execute basic and instrumental activities of daily living (ADL) and leisure activities. The scale consists of 40 questions assessing basic and instrumental ADLs. This scale assessed a participants' ability to initiate, plan, and perform activities related to hygiene, dressing, continence, eating, meal preparation, telephoning, going on an outing, finance and correspondence, medications, leisure, and housework. Each item was scored as yes: 1, no: 0 and N/A: not applicable. Higher scores indicate less disability with a score of 100 indicating no disability and 0 indicating no functional ability. The percentage score was calculated as (DAD Total score /Total number of applicable items) multiplied by 100. Change from Baseline was calculated as value at scheduled time point minus Baseline value. Baseline was defined as value at Week 0. Full population data was presented.
Time Frame: Baseline (Week 0) and Week 8, 16, 24, 48
Population: ITT population. Number of participants with observed data contributing to the analysis.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | RSG XR 2mg | RSG XR 8mg
Number analyzed (Participants) | 479 | 480 | 470
Scores on a scale
  Week 8: number analyzed (Participants) | 464 | 455 | 442
  Week 8 | -2.3 (0.50) | -1.2 (0.50) | -2.3 (0.46)
  Week 16: number analyzed (Participants) | 443 | 433 | 417
  Week 16 | -3.0 (0.57) | -2.3 (0.55) | -3.9 (0.59)
  Week 24: number analyzed (Participants) | 427 | 412 | 387
  Week 24 | -4.6 (0.60) | -2.8 (0.62) | -4.7 (0.63)
  Week 48: number analyzed (Participants) | 373 | 359 | 342
  Week 48 | -9.5 (0.81) | -9.4 (0.81) | -10.4 (0.82)
Statistical Analysis 1: Comparison: Placebo vs RSG XR 2mg; For Week 8; Test type: Superiority; p = 0.090, Mixed model for repeated measures; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Net) = 1.1, 95% CI 2-sided [-0.2 to 2.5] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs RSG XR 8mg; For Week 8; Test type: Superiority; p = 0.957, Mixed model for repeated measures; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Net) = 0.0, 95% CI 2-sided [-1.3 to 1.3] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs RSG XR 2mg; For Week 16; Test type: Superiority; p = 0.395, Mixed model for repeated measures; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Net) = 0.7, 95% CI 2-sided [-0.9 to 2.2] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Placebo vs RSG XR 8mg; For Week 16; Test type: Superiority; p = 0.275, Mixed model for repeated measures; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Net) = -0.9, 95% CI 2-sided [-2.5 to 0.7] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Placebo vs RSG XR 2mg; For Week 24; Test type: Superiority; p = 0.039, Mixed model for repeated measures; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Net) = 1.7, 95% CI 2-sided [0.1 to 3.4] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Placebo vs RSG XR 8mg; For Week 24; Test type: Superiority; p = 0.895, Mixed model for repeated measures; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Net) = -0.1, 95% CI 2-sided [-1.8 to 1.6] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: Placebo vs RSG XR 2mg; For Week 48; Test type: Superiority; p = 0.914, Mixed model for repeated measures; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Net) = 0.1, 95% CI 2-sided [-2.1 to 2.3] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 8: Comparison: Placebo vs RSG XR 8mg; For Week 48; Test type: Superiority; p = 0.430, Mixed model for repeated measures; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Net) = -0.9, 95% CI 2-sided [-3.2 to 1.3] — [estimate comment as in outcome 1, analysis 1]

11. Secondary Outcome: Change From Baseline in Neuropsychiatric Inventory (NPI) Total Score
Description: NPI is an assessment of frequency and severity of behavioral disturbances in dementia that comprised of 10 dimensions: delusions, hallucinations, dysphoria, apathy, euphoria, disinhibition, aggressiveness and agitation, irritability, anxiety, aberrant motor activity. Participant's caregiver asked about behavior in participant. If "Yes", informant then rated both severity on a 3-point scale, 1-mild to 3-severe (total range: 0-36) and frequency using a 4-point scale, 1-occasionally to 4-very frequently. Total score was frequency × severity. Distress was scored on 5-point scale, 0-no distress to 5-very severe or extreme. Total NPI score was calculated by adding all domain scores; NPI total score: 0-144 and NPI distress score: 0-60, higher scores indicated more severe behavioral disturbance. Change from Baseline was calculated as value at scheduled time point minus Baseline value. Baseline was defined as value at Week 0. Adjusted means were presented. Full population data was presented.
Time Frame: Baseline (Week 0) and Week 8, 16, 24, 48
Population: ITT population. Number of participants with observed data contributing to the analysis.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | RSG XR 2mg | RSG XR 8mg
Number analyzed (Participants) | 479 | 480 | 470
Scores on a scale
  Week 8: number analyzed (Participants) | 464 | 457 | 443
  Week 8 | -0.0 (0.32) | -0.3 (0.33) | -0.2 (0.31)
  Week 16: number analyzed (Participants) | 443 | 433 | 417
  Week 16 | 0.1 (0.34) | 0.2 (0.37) | 0.1 (0.37)
  Week 24: number analyzed (Participants) | 428 | 413 | 384
  Week 24 | 1.3 (0.43) | 0.3 (0.41) | 0.2 (0.39)
  Week 48: number analyzed (Participants) | 374 | 360 | 342
  Week 48 | 2.6 (0.52) | 1.5 (0.49) | 1.9 (0.50)
Statistical Analysis 1: Comparison: Placebo vs RSG XR 2mg; For Week 8; Test type: Superiority; p = 0.583, Mixed model for repeated measures; Mean Difference (Net) = -0.2, 95% CI 2-sided [-1.1 to 0.6]
Statistical Analysis 2: Comparison: Placebo vs RSG XR 8mg; For Week 8; Test type: Superiority; p = 0.631, Mixed model for repeated measures; Mean Difference (Net) = -0.2, 95% CI 2-sided [-1.1 to 0.6]
Statistical Analysis 3: Comparison: Placebo vs RSG XR 2mg; For Week 16; Test type: Superiority; p = 0.812, Mixed model for repeated measures; Mean Difference (Net) = 0.1, 95% CI 2-sided [-0.8 to 1.1]
Statistical Analysis 4: Comparison: Placebo vs RSG XR 8mg; For Week 16; Test type: Superiority; p = 0.952, Mixed model for repeated measures; Mean Difference (Net) = 0.0, 95% CI 2-sided [-0.9 to 1.0]
Statistical Analysis 5: Comparison: Placebo vs RSG XR 2mg; For Week 24; Test type: Superiority; p = 0.117, Mixed model for repeated measures; Mean Difference (Net) = -0.9, 95% CI 2-sided [-2.1 to 0.2]
Statistical Analysis 6: Comparison: Placebo vs RSG XR 8mg; For Week 24; Test type: Superiority; p = 0.074, Mixed model for repeated measures; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Net) = -1.0, 95% CI 2-sided [-2.1 to 0.1] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: Placebo vs RSG XR 2mg; For Week 48; Test type: Superiority; p = 0.141, Mixed model for repeated measures; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Net) = -1.0, 95% CI 2-sided [-2.4 to 0.3] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 8: Comparison: Placebo vs RSG XR 8mg; For Week 48; Test type: Superiority; p = 0.331, Mixed model for repeated measures; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Net) = -0.7, 95% CI 2-sided [-2.1 to 0.7] — [estimate comment as in outcome 1, analysis 1]

12. Secondary Outcome: Change From Baseline in Domains of the Resource Utilization in Dementia Scale (RUD)- Q1 and Q2 Caregiver Hours
Description: The RUD instrument was developed as a comprehensive tool to assess the amount of resource use among demented patients. RUD assessd both formal and informal resource use of the patient and the primary caregiver, making it possible to calculate costs from a societal perspective. Q1 corresponds to the number of hours during the last month the caregiver spent assisting the patient with toilet visits, eating, dressing, grooming, walking and bathing and Q2 corresponds to the number of hours during the last month the caregiver spent assisting the patient with shopping, food preparation, housekeeping, laundry, transportation, taking medication and managing financial matters. Change from Baseline was calculated as value at scheduled time point minus Baseline value. Baseline was defined as value at Week 0. Estimated value was calculated by Active treatment minus Placebo. The adjusted means were presented. Full population data was presented.
Time Frame: Baseline (Week 0) and Week 12, 24, 36, 48
Population: ITT population. Number of participants with observed data contributing to the analysis.
Measure: Least Squares Mean (Standard Error); unit: Caregiver hours
Arm/Group | Placebo | RSG XR 2mg | RSG XR 8mg
Number analyzed (Participants) | 479 | 480 | 470
Caregiver hours
  Q1 Week 12: number analyzed (Participants) | 449 | 441 | 425
  Q1 Week 12 | -2.4 (2.72) | 1.8 (2.56) | 3.5 (2.68)
  Q1 Week 24: number analyzed (Participants) | 427 | 411 | 385
  Q1 Week 24 | 7.4 (3.43) | 9.0 (2.92) | 10.9 (3.69)
  Q1 Week 36: number analyzed (Participants) | 393 | 383 | 359
  Q1 Week 36 | 11.2 (4.36) | 12.7 (3.70) | 13.4 (4.09)
  Q1 Week 48: number analyzed (Participants) | 371 | 357 | 341
  Q1 Week 48 | 15.7 (4.14) | 19.7 (4.06) | 19.2 (4.54)
  Q2 Week 12: number analyzed (Participants) | 448 | 440 | 425
  Q2 Week 12 | -1.1 (4.06) | 5.8 (3.70) | 6.4 (4.04)
  Q2 Week 24: number analyzed (Participants) | 427 | 410 | 385
  Q2 Week 24 | 5.6 (4.41) | 15.6 (4.90) | 12.3 (4.79)
  Q2 Week 36: number analyzed (Participants) | 393 | 382 | 359
  Q2 Week 36 | 16.4 (5.52) | 23.4 (6.10) | 15.2 (4.53)
  Q2 Week 48: number analyzed (Participants) | 371 | 356 | 341
  Q2 Week 48 | 21.8 (5.62) | 26.0 (5.69) | 21.6 (4.92)
Statistical Analysis 1: Comparison: Placebo vs RSG XR 2mg; Q1 Week 12; Test type: Superiority; p = 0.251, Mixed model for repeated measures; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Net) = 4.1, 95% CI 2-sided [-2.9 to 11.2] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs RSG XR 8mg; Q1 Week 12; Test type: Superiority; p = 0.113, Mixed model for repeated measures; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Net) = 5.9, 95% CI 2-sided [-1.4 to 13.2] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs RSG XR 2mg; Q1 Week 24; Test type: Superiority; p = 0.723, Mixed model for repeated measures; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Net) = 1.6, 95% CI 2-sided [-7.1 to 10.2] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Placebo vs RSG XR 8mg; Q1 Week 24; Test type: Superiority; p = 0.482, Mixed model for repeated measures; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Net) = 3.5, 95% CI 2-sided [-6.3 to 13.2] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Placebo vs RSG XR 2mg; Q1 Week 36; Test type: Superiority; p = 0.785, Mixed model for repeated measures; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Net) = 1.5, 95% CI 2-sided [-9.5 to 12.6] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Placebo vs RSG XR 8mg; Q1 Week 36; Test type: Superiority; p = 0.711, Mixed model for repeated measures; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Net) = 2.2, 95% CI 2-sided [-9.4 to 13.8] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: Placebo vs RSG XR 2mg; Q1 Week 48; Test type: Superiority; p = 0.484, Mixed model for repeated measures; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Net) = 4.0, 95% CI 2-sided [-7.2 to 15.2] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 8: Comparison: Placebo vs RSG XR 8mg; Q1 Week 48; Test type: Superiority; p = 0.572, Mixed model for repeated measures; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Net) = 3.4, 95% CI 2-sided [-8.5 to 15.4] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 9: Comparison: Placebo vs RSG XR 2mg; Q2 Week 12; Test type: Superiority; p = 0.197, Mixed model for repeated measures; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Net) = 6.8, 95% CI 2-sided [-3.6 to 17.3] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 10: Comparison: Placebo vs RSG XR 8mg; Q2 Week 12; Test type: Superiority; p = 0.183, Mixed model for repeated measures; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Net) = 7.4, 95% CI 2-sided [-3.5 to 18.4] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 11: Comparison: Placebo vs RSG XR 2mg; Q2 Week 24; Test type: Superiority; p = 0.121, Mixed model for repeated measures; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Net) = 10.0, 95% CI 2-sided [-2.6 to 22.6] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 12: Comparison: Placebo vs RSG XR 8mg; Q2 Week 24; Test type: Superiority; p = 0.291, Mixed model for repeated measures; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Net) = 6.8, 95% CI 2-sided [-5.8 to 19.3] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 13: Comparison: Placebo vs RSG XR 2mg; Q2 Week 36; Test type: Superiority; p = 0.389, Mixed model for repeated measures; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Net) = 7.0, 95% CI 2-sided [-8.9 to 22.9] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 14: Comparison: Placebo vs RSG XR 8mg; Q2 Week 36; Test type: Superiority; p = 0.865, Mixed model for repeated measures; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Net) = -1.2, 95% CI 2-sided [-15.0 to 12.6] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 15: Comparison: Placebo vs RSG XR 2mg; Q2 Week 48; Test type: Superiority; p = 0.596, Mixed model for repeated measures; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Net) = 4.2, 95% CI 2-sided [-11.3 to 19.6] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 16: Comparison: Placebo vs RSG XR 8mg; Q2 Week 48; Test type: Superiority; p = 0.975, Mixed model for repeated measures; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Net) = -0.2, 95% CI 2-sided [-14.7 to 14.2] — [estimate comment as in outcome 1, analysis 1]

13. Secondary Outcome: Change From Baseline in European Quality of Life -5 Dimensions (EQ-5D) Scale Total Score- Thermometer Score
Description: The EQ-5D Proxy is an assessment of quality of life and utility benefit. The EQ-5D Proxy is composed of two parts: part two is the visual analogue scale 'Thermometer'. Caregivers are asked to respond as they feel the participant would on dimensions of mobility, self-care, usual activities, pain/discomfort and anxiety/depression. The 'Thermometer' has endpoints of 100 (best imaginable health state) and 0 (worst imaginable health state). Change from Baseline was calculated as value at scheduled time point minus Baseline value. Baseline was defined as value a t Week 0. Estimated value was calculated by Active treatment minus Placebo. The adjusted means were presented. Full population data was presented.
Time Frame: Baseline (Week 0) and Week 12, 36, 48
Population: ITT population. Number of participants with observed data contributing to the analysis.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | RSG XR 2mg | RSG XR 8mg
Number analyzed (Participants) | 479 | 480 | 470
Scores on a scale
  Thermometer score Week 12: number analyzed (Participants) | 442 | 439 | 424
  Thermometer score Week 12 | 2.4 (0.82) | -0.0 (0.89) | 0.1 (0.87)
  Thermometer score Week 36: number analyzed (Participants) | 396 | 383 | 361
  Thermometer score Week 36 | 1.7 (0.87) | 1.3 (0.94) | -0.4 (0.95)
  Thermometer score Week 48: number analyzed (Participants) | 366 | 354 | 342
  Thermometer score Week 48 | 2.1 (0.91) | -0.5 (1.00) | -1.4 (0.96)
Statistical Analysis 1: Comparison: Placebo vs RSG XR 2mg; Thermometer score Week 12; Test type: Superiority; p = 0.043, Mixed model for repeated measures; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Net) = -2.4, 95% CI 2-sided [-4.7 to -0.1] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs RSG XR 8mg; Thermometer score Week 12; Test type: Superiority; p = 0.056, Mixed model for repeated measures; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Net) = -2.2, 95% CI 2-sided [-4.5 to 0.1] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs RSG XR 2mg; Thermometer score Week 36; Test type: Superiority; p = 0.758, Mixed model for repeated measures; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Net) = -0.4, 95% CI 2-sided [-2.8 to 2.1] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Placebo vs RSG XR 8mg; Thermometer score Week 36; Test type: Superiority; p = 0.109, Mixed model for repeated measures; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Net) = -2.0, 95% CI 2-sided [-4.5 to 0.5] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Placebo vs RSG XR 2mg; Thermometer score Week 48; Test type: Superiority; p = 0.050, Mixed model for repeated measures; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Net) = -2.6, 95% CI 2-sided [-5.2 to -0.0] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Placebo vs RSG XR 8mg; Thermometer score Week 48; Test type: Superiority; p = 0.009, Mixed model for repeated measures; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Net) = -3.4, 95% CI 2-sided [-6.0 to -0.9] — [estimate comment as in outcome 1, analysis 1]

14. Secondary Outcome: Change From Baseline in EQ-5D Scale Total Score- Utility Score
Description: The EQ-5D Proxy is an assessment of quality of life and utility benefit. The EQ-5D Proxy is composed of two parts: part one is the five dimensional Health State Classification. The Utility score is a caregiver rating of health status on dimensions of mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Answers to each question were responded to on a 3-point scale which indicates the level of impairment (level 1= no problem; level 2=some or moderate problem(s) and level 3=unable, or extreme problem with higher scores indicating greater dysfunction. Change from Baseline was calculated as value at scheduled time point minus Baseline value. Baseline was defined as value a t Week 0. Estimated value was calculated by Active treatment minus Placebo. The adjusted means were presented. Full population data was presented.
Time Frame: Baseline (Week 0) and Week 12, 36, 48
Population: ITT population. Number of participants with observed data contributing to the analysis.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | RSG XR 2mg | RSG XR 8mg
Number analyzed (Participants) | 479 | 480 | 470
Scores on a scale
  Ultility score Week 12: number analyzed (Participants) | 442 | 441 | 423
  Ultility score Week 12 | -0.02 (0.009) | -0.01 (0.009) | -0.03 (0.009)
  Utility score Week 36: number analyzed (Participants) | 397 | 385 | 362
  Utility score Week 36 | -0.03 (0.011) | -0.03 (0.011) | -0.06 (0.010)
  Utility score Week 48: number analyzed (Participants) | 368 | 355 | 342
  Utility score Week 48 | -0.03 (0.011) | -0.05 (0.012) | -0.04 (0.010)
Statistical Analysis 1: Comparison: Placebo vs RSG XR 2mg; Ultility score Week 12; Test type: Superiority; p = 0.662, Mixed model for repeated measures; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Net) = 0.01, 95% CI 2-sided [-0.02 to 0.03] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs RSG XR 8mg; Ultility score Week 12; Test type: Superiority; p = 0.503, Mixed model for repeated measures; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Net) = -0.01, 95% CI 2-sided [-0.03 to 0.02] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs RSG XR 2mg; Utility score Week 36; Test type: Superiority; p = 0.892, Mixed model for repeated measures; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Net) = 0.00, 95% CI 2-sided [-0.03 to 0.03] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Placebo vs RSG XR 8mg; Utility score Week 36; Test type: Superiority; p = 0.083, Mixed model for repeated measures; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Net) = -0.03, 95% CI 2-sided [-0.05 to 0.00] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Placebo vs RSG XR 2mg; Utility score Week 48; Test type: Superiority; p = 0.366, Mixed model for repeated measures; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Net) = -0.01, 95% CI 2-sided [-0.05 to 0.02] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Placebo vs RSG XR 8mg; Utility score Week 48; Test type: Superiority; p = 0.769, Mixed model for repeated measures; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Net) = -0.00, 95% CI 2-sided [-0.03 to 0.02] — [estimate comment as in outcome 1, analysis 1]

15. Secondary Outcome: Change From Baseline in Alzheimer's Carer's Quality of Life Instrument (ACQLI) Score
Description: The ACQLI is an assessment of caregiver quality of life. This instrument consisted of 30 questions exploring various aspects of carer's quality of life. Each of the questions had two point response, and the 30 questions were summed to provide a total score. Items were assumed to be unidimensional (i.e., represent a single variable) and were scored 0/1 (false/true) before summation into a total score with a 0-30 range. To ease comparisons between scales, ACQLI scores were transformed to range between 0-100 (100: worse). Change from Baseline was calculated as value at scheduled time point minus Baseline value. Baseline was defined as value a t Week 0. Estimated value was calculated by Active treatment minus Placebo. The adjusted means were presented. Full population data was presented.
Time Frame: Baseline (Week 0) and Week 12, 36, 48
Population: ITT population. Number of participants with observed data contributing to the analysis.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | RSG XR 2mg | RSG XR 8mg
Number analyzed (Participants) | 479 | 480 | 470
Scores on a scale
  Week 12: number analyzed (Participants) | 447 | 443 | 419
  Week 12 | 0.3 (0.19) | 0.1 (0.19) | 0.2 (0.21)
  Week 36: number analyzed (Participants) | 400 | 384 | 361
  Week 36 | 1.2 (0.24) | 0.8 (0.25) | 1.4 (0.25)
  Week 48: number analyzed (Participants) | 373 | 356 | 341
  Week 48 | 1.1 (0.27) | 1.3 (0.29) | 1.2 (0.27)
Statistical Analysis 1: Comparison: Placebo vs RSG XR 2mg; Week 12; Test type: Superiority; p = 0.529, Mixed model for repeated measures; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Net) = -0.2, 95% CI 2-sided [-0.7 to 0.3] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs RSG XR 8mg; Week 12; Test type: Superiority; p = 0.620, Mixed model for repeated measures; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Net) = -0.1, 95% CI 2-sided [-0.7 to 0.4] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs RSG XR 2mg; Week 36; Test type: Superiority; p = 0.284, Mixed model for repeated measures; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Net) = -0.4, 95% CI 2-sided [-1.0 to 0.3] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Placebo vs RSG XR 8mg; Week 36; Test type: Superiority; p = 0.488, Mixed model for repeated measures; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Net) = 0.2, 95% CI 2-sided [-0.4 to 0.9] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Placebo vs RSG XR 2mg; Week 48; Test type: Superiority; p = 0.549, Mixed model for repeated measures; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Net) = 0.2, 95% CI 2-sided [-0.5 to 1.0] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Placebo vs RSG XR 8mg; For Week 48; Test type: Superiority; p = 0.780, Mixed model for repeated measures; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Net) = 0.1, 95% CI 2-sided [-0.6 to 0.9] — [estimate comment as in outcome 1, analysis 1]

16. Secondary Outcome: Change in ADAS-Cog Total Score for Observed Cases at Week 54 Compared to Week 48
Description: The 11-item ADAS-Cog assessed a range of cognitive abilities including memory, comprehension, orientation in time and place and spontaneous speech. Most items were evaluated by tests, but some were dependent on clinician ratings on a five point scale. Scores range from 0 to 70 with higher scores indicating greater dysfunction. It was of interest to compare the single blind phase data between the treatment groups defined based on the double blind treatment group. This analysis only included participants who received at least one dose of single-blind medication. Change from Baseline was calculated as value at scheduled time point minus Baseline value. Baseline was defined as value at Week 0. Full population data was presented.
Time Frame: Week 48 and Week 54
Population: ITT population. This analysis will only include participants who received at least one dose of single-blind medication. Only those participants available at that particular time point were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | RSG XR 2mg | RSG XR 8mg
Number analyzed (Participants) | 338 | 319 | 307
Scores on a scale | 1.0 (0.27) | 0.4 (0.28) | 0.5 (0.28)
Statistical Analysis 1: Comparison: Placebo vs RSG XR 2mg; Test type: Superiority; p = 0.106, ANCOVA; Mean Difference (Net) = -0.6, 95% CI 2-sided [-1.3 to 0.1]
Statistical Analysis 2: Comparison: Placebo vs RSG XR 8mg; Test type: Superiority; p = 0.229, ANCOVA; Mean Difference (Net) = -0.4, 95% CI 2-sided [-1.2 to 0.3]

17. Secondary Outcome: Change in CDR-SB Total Score for Observed Cases at Week 54 Compared to Week 48
Description: The CDR-SB was a validated clinical assessment of global function in participants with AD. Impairment was scored in each of 6 cognitive categories on a scale in which none = 0, questionable = 0.5, mild = 1, moderate = 2, and severe = 3. The 6 individual category ratings, or "box scores", can be added together to give the CDR-Sum of Boxes which ranges from 0 to 18 (severe impairment). It was of interest to compare the single blind phase data between the treatment groups defined based on the double blind treatment group. This analysis only included participants who received at least one dose of single-blind medication. Change from Baseline was calculated as value at scheduled time point minus Baseline value. Baseline was defined as value at Week 0. Full population data was presented.
Time Frame: Week 48 and Week 54
Population: ITT population. Only those participants available at that particular time point were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | RSG XR 2mg | RSG XR 8mg
Number analyzed (Participants) | 335 | 316 | 303
Scores on a scale | 0.3 (0.07) | 0.2 (0.08) | 0.3 (0.08)
Statistical Analysis 1: Comparison: Placebo vs RSG XR 2mg; Test type: Superiority; p = 0.324, ANCOVA; Mean Difference (Net) = -0.1, 95% CI 2-sided [-0.3 to 0.1]
Statistical Analysis 2: Comparison: Placebo vs RSG XR 8mg; Test type: Superiority; p = 0.987, ANCOVA; Mean Difference (Net) = 0.0, 95% CI 2-sided [-0.2 to 0.2]

18. Secondary Outcome: Change From Baseline in Glycosylated Hemoglobin (HbA1c) at Week 48
Description: Blood samples were collected for assessments of HbA1c levels at Baseline and up to Week 48. Change from Baseline was calculated as value at scheduled time point minus Baseline value . Baseline was defined as value at Week 0. Endpoint treatment differences which were adjusted to take account of missing data are derived. Full population data was presented.
Time Frame: Baseline (Week 0) and Week 48
Population: ITT population. Only those participants available at that particular time point were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Percentage
Arm/Group | Placebo | RSG XR 2mg | RSG XR 8mg
Number analyzed (Participants) | 337 | 326 | 309
Percentage | 0.13 (0.018) | 0.18 (0.019) | 0.26 (0.019)
Statistical Analysis 1: Comparison: Placebo vs RSG XR 2mg; Test type: Superiority; p = 0.038, ANCOVA; Mean Difference (Net) = 0.05, 95% CI 2-sided [0.00 to 0.10]
Statistical Analysis 2: Comparison: Placebo vs RSG XR 8mg; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Net) = 0.13, 95% CI 2-sided [0.08 to 0.18]

19. Secondary Outcome: Number of Participants With On-treatment Adverse Events (AEs), Serious Adverse Events (SAEs) and Severity of AEs
Description: AE was defined as any untoward medical occurrence in a participant temporarily associated with the use of a medicinal product, whether or not considered related to the medicinal product. SAE was any untoward medical occurrence that, at any dose results in death, was life threatening, required hospitalization or prolongation of existing hospitalization, resulted in disability/incapacity, was a congenital anomaly/birth defect or was considered as medically significant.
Time Frame: Upto Week 48
Population: Safety population consisted of all participants randomized to treatment who had taken at least one dose of study medication. This population was used for analysis of safety data.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | RSG XR 2mg | RSG XR 8mg
Number analyzed (Participants) | 487 | 490 | 491
Participants
  On treatment AEs | 275 | 298 | 319
  On treatment SAEs | 60 | 58 | 66
  Mild AEs | 109 | 119 | 112
  Moderate AEs | 111 | 128 | 158
  Severe AEs | 55 | 50 | 48

20. Secondary Outcome: Number of Participants With Change From Baseline in Vital Signs of Clinical Concern at Any Time on Treatment- Weight
Description: Body weight was measured at all visits, without shoes and wearing light clothing. The assessment was performed a t Baseline and up to Week 54. Change from Baseline was calculated as value at scheduled time point minus Baseline value. Baseline was defined as value at Week 0. Full population data was presented.
Time Frame: Upto Week 54
Population: Safety population. Only those participants available at the indicated time point were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | RSG XR 2mg | RSG XR 8mg
Number analyzed (Participants) | 355 | 342 | 318
Participants
  Increase from Baseline >=7% | 33 | 31 | 47
  Decrease from Baseline >=7% | 28 | 32 | 23

21. Secondary Outcome: Number of Participants With Change From Baseline in Vital Signs of Clinical Concern at Any Time on Treatment- Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP)
Description: SBP and DBP of participants were recorded in sitting posture as vital sign at each visit. The blood pressure (BP) values were identified as of potential clinical concern if the values were out of the reference range (for SBP, 90 to 140 mmHg and DBP, 50 to 90 mmHg) or meet a change from baseline criterion. The change from baseline criterion for SBP, was increase from Baseline (high) if increased by more than or equal to (>=) 40 mm Hg from Baseline; decrease from Baseline (low) if decreased by >= 30 mmHg from Baseline. For DBP, increase from baseline (high) if increased by >=30 mmHg from baseline; decrease from Baseline (low) if decreased by >= 20 mmHg from Baseline. Baseline was defined as value at Week 0.
Time Frame: Upto Week 54
Population: Safety population. Only those participants available at the indicated time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | RSG XR 2mg | RSG XR 8mg
Number analyzed (Participants) | 487 | 490 | 491
Participants
  SBP >140 or <90: number analyzed (Participants) | 356 | 343 | 322
  SBP >140 or <90 | 67 | 72 | 86
  SBP Increase from Baseline>=40: number analyzed (Participants) | 356 | 343 | 322
  SBP Increase from Baseline>=40 | 1 | 3 | 3
  SBP Decrease from Baseline>=30: number analyzed (Participants) | 356 | 343 | 322
  SBP Decrease from Baseline>=30 | 19 | 19 | 14
  DBP >90 or <50: number analyzed (Participants) | 356 | 343 | 322
  DBP >90 or <50 | 8 | 15 | 12
  DBP Increase from Baseline>=30: number analyzed (Participants) | 356 | 343 | 322
  DBP Increase from Baseline>=30 | 0 | 0 | 1
  DBP Decrease from Baseline >=20: number analyzed (Participants) | 356 | 343 | 322
  DBP Decrease from Baseline >=20 | 12 | 18 | 13

22. Secondary Outcome: Number of Participants With Change From Baseline in Vital Signs of Clinical Concern at Any Time on Treatment- Heart Rate (HR)
Description: HR of participants were recorded in sitting posture as vital sign at each visit. The HR values were identified as of potential clinical concern if the values were out of the reference range (50 to 100 beats per minute) or meet a change from baseline criterion. The change from baseline criterion for HR, was increase from Baseline (high) if increased by more than or equal to (>=) 30 from Baseline; decrease from Baseline (low) if decreased by >= 30 from Baseline. Baseline was defined as value at Week 0. Full population data was presented.
Time Frame: Upto Week 54
Population: Safety population. Only those participants available at the indicated time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | RSG XR 2mg | RSG XR 8mg
Number analyzed (Participants) | 355 | 344 | 322
Participants
  >100 or <50 | 12 | 5 | 5
  Increase from Baseline >=30 | 0 | 0 | 4
  Decrease from Baseline >=30 | 2 | 0 | 1

23. Secondary Outcome: Change From Baseline in Weight
Description: Body weight was measured at all visits, without shoes and wearing light clothing. The assessment was performed at Baseline, Weeks 4, 8, 12, 16, 24, 36, 48, 54. Change from Baseline was calculated as value at scheduled time point minus Baseline value. Baseline was defined as value at Week 0. Full population data was presented.
Time Frame: Baseline (Week 0) and Weeks 4, 8, 12, 16, 24, 36, 48, 54
Population: Safety population. Only those participants available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Kilograms (Kg)
Arm/Group | Placebo | RSG XR 2mg | RSG XR 8mg
Number analyzed (Participants) | 487 | 490 | 491
Kilograms (Kg)
  Week 4: number analyzed (Participants) | 470 | 471 | 469
  Week 4 | -0.1 (1.95) | 0.1 (1.61) | 0.5 (1.70)
  Week 8: number analyzed (Participants) | 459 | 447 | 443
  Week 8 | 0.1 (2.10) | 0.2 (2.15) | 0.9 (2.34)
  Week 12: number analyzed (Participants) | 447 | 436 | 420
  Week 12 | 0.0 (2.35) | 0.1 (2.66) | 1.2 (2.50)
  Week 16: number analyzed (Participants) | 440 | 428 | 416
  Week 16 | 0.0 (2.88) | 0.2 (2.85) | 1.3 (2.78)
  Week 24: number analyzed (Participants) | 428 | 412 | 387
  Week 24 | 0.1 (2.85) | 0.1 (3.28) | 1.2 (3.59)
  Week 36: number analyzed (Participants) | 397 | 389 | 359
  Week 36 | -0.0 (4.53) | 0.2 (3.69) | 1.5 (3.28)
  Week 48: number analyzed (Participants) | 375 | 358 | 341
  Week 48 | 0.1 (3.51) | 0.2 (4.33) | 1.9 (3.69)
  Week 54: number analyzed (Participants) | 355 | 342 | 318
  Week 54 | 0.1 (3.70) | 0.1 (5.88) | 1.2 (3.57)

24. Secondary Outcome: Change From Baseline in Hemoglobin
Description: Hematology parameters were assessed at Baseline, Weeks 4, 16, 36, 48. Change from Baseline was calculated as value at scheduled time point minus Baseline value. Baseline was defined as value at Week 0. Full population data was presented.
Time Frame: Baseline (Week 0) and Weeks 4, 16, 36, 48
Population: Safety population. Only those participants available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Gram\Liter (G\L)
Arm/Group | Placebo | RSG XR 2mg | RSG XR 8mg
Number analyzed (Participants) | 487 | 490 | 491
Gram\Liter (G\L)
  Week 4: number analyzed (Participants) | 460 | 453 | 461
  Week 4 | -0.5 (6.50) | -2.9 (6.76) | -3.9 (6.80)
  Week 16: number analyzed (Participants) | 428 | 422 | 403
  Week 16 | -0.6 (7.37) | -6.1 (7.79) | -11.2 (9.37)
  Week 36: number analyzed (Participants) | 381 | 376 | 343
  Week 36 | -0.7 (7.78) | -6.2 (8.73) | -10.6 (9.67)
  Week 48: number analyzed (Participants) | 362 | 336 | 332
  Week 48 | -0.7 (9.10) | -5.8 (8.66) | -10.7 (10.15)

25. Secondary Outcome: Change From Baseline in Hematocrit
Description: Hematology parameters were assessed at Baseline and up to Week 48. Change from Baseline was calculated as value at scheduled time point minus Baseline value. Baseline was defined as value at Week 0.
Time Frame: Baseline (Week 0) and Weeks 4, 16, 36, 48
Population: Safety population. Only those participants available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Placebo | RSG XR 2mg | RSG XR 8mg
Number analyzed (Participants) | 487 | 490 | 491
Ratio
  Week 4: number analyzed (Participants) | 459 | 453 | 461
  Week 4 | -0.0020 (0.02050) | -0.0088 (0.02150) | -0.0121 (0.02128)
  Week 16: number analyzed (Participants) | 428 | 422 | 403
  Week 16 | -0.0018 (0.02340) | -0.0166 (0.02442) | -0.0320 (0.02922)
  Week 36: number analyzed (Participants) | 381 | 376 | 343
  Week 36 | -0.0017 (0.02428) | -0.0174 (0.02705) | -0.0300 (0.02880)
  Week 48: number analyzed (Participants) | 362 | 336 | 332
  Week 48 | -0.0026 (0.02776) | -0.0167 (0.02683) | -0.0303 (0.03015)

26. Secondary Outcome: Any Time on Treatment Differences in Frequencies of Hematology Data Outside the Reference Range
Description: Haematology parameters were identified as of PCC (high [H], low [L]), if the values were out of the reference range (RR). The range for parameters was: platelet (100AV-500AV), red blood cell (RBC , 0.8-1.2), hemoglobin (L: female [F]:10, male [M]:11; H: F:16.5-AV, M:18), hematocrit (0.8-1.2), white blood cell (WBC, 3-15), Total neutrophils (ANC- absolute Neutrophil count) (0.75-1.5), lymphocytes (0.75-1.5), monocyte s (0.75-2), eosinophils (none -2), basophils (none -2), mean corpuscle volume (MCV, 0.8-1.2), mean corpuscular hemoglobin (MCH, 0.8-1.2), mean corpuscular hemoglobin concentration (MCHC , 0.8-1.2), red cell distribution width (RDW, 0.8-1.2), Neutrophil bands (none-1) and segmented neutrophils (0.75-1.3). Full population data was presented.
Time Frame: Up to Week 48
Population: Safety population. Only those participants available at the indicated time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | RSG XR 2mg | RSG XR 8mg
Number analyzed (Participants) | 487 | 490 | 491
Participants
  Eosinophils- High: number analyzed (Participants) | 474 | 473 | 472
  Eosinophils- High | 3 | 1 | 1
  Hematocrit- Low: number analyzed (Participants) | 474 | 473 | 472
  Hematocrit- Low | 3 | 3 | 6
  Hemoglobin- High: number analyzed (Participants) | 474 | 473 | 474
  Hemoglobin- High | 1 | 3 | 1
  Hemoglobin- Low: number analyzed (Participants) | 474 | 473 | 472
  Hemoglobin- Low | 9 | 14 | 36
  Lymphocytes- High: number analyzed (Participants) | 474 | 473 | 472
  Lymphocytes- High | 3 | 1 | 1
  Lymphocytes- Low: number analyzed (Participants) | 474 | 473 | 472
  Lymphocytes- Low | 11 | 3 | 7
  MCH- High: number analyzed (Participants) | 474 | 473 | 472
  MCH- High | 0 | 0 | 1
  MCH- Low: number analyzed (Participants) | 474 | 473 | 472
  MCH- Low | 1 | 3 | 3
  MCV- High: number analyzed (Participants) | 474 | 473 | 472
  MCV- High | 0 | 0 | 1
  MCV- Low: number analyzed (Participants) | 474 | 473 | 472
  MCV- Low | 0 | 1 | 1
  Monocytes- Low: number analyzed (Participants) | 474 | 473 | 472
  Monocytes- Low | 44 | 21 | 44
  Platelet count- High: number analyzed (Participants) | 475 | 473 | 472
  Platelet count- High | 3 | 2 | 4
  Platelet count- Low: number analyzed (Participants) | 475 | 473 | 472
  Platelet count- Low | 3 | 0 | 2
  RDW- High: number analyzed (Participants) | 474 | 474 | 472
  RDW- High | 11 | 18 | 50
  RDW- Low: number analyzed (Participants) | 474 | 474 | 472
  RDW- Low | 1 | 0 | 0
  Red Blood Cell count- High: number analyzed (Participants) | 474 | 473 | 472
  Red Blood Cell count- High | 0 | 0 | 1
  Red Blood Cell count- Low: number analyzed (Participants) | 474 | 473 | 472
  Red Blood Cell count- Low | 3 | 3 | 11
  Total Neutrophils (ANC)- High: number analyzed (Participants) | 474 | 473 | 472
  Total Neutrophils (ANC)- High | 4 | 0 | 0
  Total Neutrophils (ANC)- Low: number analyzed (Participants) | 474 | 473 | 472
  Total Neutrophils (ANC)- Low | 4 | 2 | 10
  White Blood Cell count- High: number analyzed (Participants) | 474 | 473 | 472
  White Blood Cell count- High | 5 | 2 | 0
  White Blood Cell count- Low: number analyzed (Participants) | 474 | 473 | 472
  White Blood Cell count- Low | 4 | 3 | 12

27. Secondary Outcome: Any Time on Treatment Differences in Frequencies of Clinical Chemistry Data Outside the Reference Range
Description: Clinical chemistry parameters were identified as of PCC (High, Low), if values were out of RR: Alanine amino transferase (ALT,none-120 [250percent upper limit of RR, ULRR ]),Album in (0.75-2),Aldolase(1.1-1.1),Aspartate amino transferase (AST,none-105 (3-64y),137.5(65+y),>250 percent ULRR), Alkaline phosphatase(ALP,none-312.5 (20+y),>250percent ULRR),blood urea nitrogen(BUN)/Creatinine ratio(none-1.25),BUN(none-11),Chloride(80-115),Calcium (0.75-1.25),Carbon dioxide(CO2,15-40) content,Creatinine (22,<50percent lower limit of RR [LLRR ]-155, >125percent ULRR),Creatine phosphokinase(CPK,none-1.25),Gamma glutamyl transferase(GGT,none-2.5),Glucose (3.6-7.8),HbA1C, High density lipoprotein (HDL,0.65-none),Lactate dehydrogenase (LDH,none -2), Low density lipoprotein(LDL,none-1.25),Magnesium (0.5-2),Potassium (3-5.5),Phosphorus inorganic(0.5-1.5), Sodium (130-150), Total protein (0.8-1.5),Total cholesterol(none -1.5),Direct Billirubin.
Time Frame: Upto Week 48
Population: Safety population. Only those participants available at the indicated time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | RSG XR 2mg | RSG XR 8mg
Number analyzed (Participants) | 487 | 490 | 491
Participants
  ALT- High: number analyzed (Participants) | 475 | 474 | 472
  ALT- High | 2 | 1 | 1
  Aldolase- High: number analyzed (Participants) | 24 | 23 | 20
  Aldolase- High | 2 | 2 | 0
  Aldolase- Low: number analyzed (Participants) | 24 | 23 | 20
  Aldolase- Low | 2 | 1 | 0
  Alkaline Phosphatase- High: number analyzed (Participants) | 475 | 474 | 472
  Alkaline Phosphatase- High | 2 | 0 | 0
  AST- High: number analyzed (Participants) | 474 | 474 | 472
  AST- High | 1 | 1 | 2
  BUN/Creatinine ratio- High: number analyzed (Participants) | 475 | 474 | 472
  BUN/Creatinine ratio- High | 17 | 25 | 40
  Calcium- Low: number analyzed (Participants) | 474 | 474 | 472
  Calcium- Low | 1 | 0 | 0
  Carbondioxide content/BicarbonateLow: number analyzed (Participants) | 474 | 474 | 472
  Carbondioxide content/BicarbonateLow | 0 | 0 | 3
  Cholesterol- High: number analyzed (Participants) | 436 | 425 | 403
  Cholesterol- High | 21 | 32 | 61
  Creatine Kinase- High: number analyzed (Participants) | 475 | 474 | 472
  Creatine Kinase- High | 33 | 63 | 69
  Creatinine- High: number analyzed (Participants) | 475 | 474 | 472
  Creatinine- High | 10 | 12 | 15
  Direct Bilirubin- High: number analyzed (Participants) | 475 | 474 | 472
  Direct Bilirubin- High | 1 | 0 | 1
  GGT- High: number analyzed (Participants) | 475 | 474 | 472
  GGT- High | 6 | 2 | 5
  Glucose- High: number analyzed (Participants) | 475 | 474 | 472
  Glucose- High | 81 | 60 | 55
  Glucose- Low: number analyzed (Participants) | 475 | 474 | 472
  Glucose- Low | 14 | 22 | 22
  Glycosylated Hemoglobin A1C: number analyzed (Participants) | 395 | 374 | 364
  Glycosylated Hemoglobin A1C | 1 | 1 | 0
  HDL Cholesterol, direct- Low: number analyzed (Participants) | 436 | 425 | 403
  HDL Cholesterol, direct- Low | 0 | 0 | 3
  LDL Cholesterol calculation- High: number analyzed (Participants) | 434 | 418 | 399
  LDL Cholesterol calculation- High | 65 | 106 | 162
  Lactate Dehydrogenase- High: number analyzed (Participants) | 474 | 474 | 472
  Lactate Dehydrogenase- High | 0 | 0 | 1
  Magnesium- Low: number analyzed (Participants) | 475 | 474 | 472
  Magnesium- Low | 1 | 0 | 1
  Phosphorus, inorganic- High: number analyzed (Participants) | 475 | 474 | 472
  Phosphorus, inorganic- High | 2 | 0 | 0
  Potassium- High: number analyzed (Participants) | 474 | 474 | 472
  Potassium- High | 11 | 12 | 12
  Potassium- Low: number analyzed (Participants) | 474 | 474 | 472
  Potassium- Low | 3 | 1 | 0
  Sodium- High: number analyzed (Participants) | 475 | 474 | 472
  Sodium- High | 2 | 0 | 2
  Sodium- Low: number analyzed (Participants) | 475 | 474 | 472
  Sodium- Low | 4 | 6 | 2
  Total Bilirubin- High: number analyzed (Participants) | 475 | 474 | 472
  Total Bilirubin- High | 5 | 1 | 1
  Troponin I- High: number analyzed (Participants) | 21 | 22 | 21
  Troponin I- High | 1 | 1 | 1
  Urea/BUN- High: number analyzed (Participants) | 475 | 474 | 472
  Urea/BUN- High | 27 | 40 | 48

28. Secondary Outcome: Changes From Baseline in Electrocardiogram (ECG) Parameters- HR
Description: Triplicate 12-lead ECG measures was obtained digitally, approximately one minute apart after the participant had rested in the supine position in a quiet room (no TV, minimal talking) for atleast 10 minutes. The ECG parameters includes HR. The assessments were performed at Baseline and up to Week 54. Change from Baseline was calculated as value at scheduled time point minus Baseline value . Baseline was defined as value at Week 0. Full population data was presented.
Time Frame: Baseline (Week 0) and Weeks 4, 8, 16, 24, 36, 48, 54
Population: Safety population. Only those participants available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Beats per minute (BPM)
Arm/Group | Placebo | RSG XR 2mg | RSG XR 8mg
Number analyzed (Participants) | 487 | 490 | 491
Beats per minute (BPM)
  Week 0, +1hr: number analyzed (Participants) | 455 | 469 | 469
  Week 0, +1hr | -1.6 (6.20) | -1.1 (5.80) | -1.8 (6.05)
  Week 0, +2hr: number analyzed (Participants) | 362 | 378 | 383
  Week 0, +2hr | -1.4 (7.05) | -0.5 (6.88) | -1.0 (7.33)
  Week 0, +3hr: number analyzed (Participants) | 229 | 234 | 246
  Week 0, +3hr | 0.0 (6.84) | -0.1 (7.02) | 0.1 (7.49)
  Week 0, +4hr: number analyzed (Participants) | 163 | 145 | 155
  Week 0, +4hr | 0.6 (6.64) | 1.0 (6.29) | 0.4 (7.84)
  Week 4, Pre-dose: number analyzed (Participants) | 443 | 442 | 443
  Week 4, Pre-dose | 0.2 (7.01) | 0.7 (7.73) | 1.0 (7.56)
  Week 4, +1hr: number analyzed (Participants) | 429 | 435 | 437
  Week 4, +1hr | -1.4 (7.98) | -0.4 (8.14) | -0.1 (7.92)
  Week 4, +2hr: number analyzed (Participants) | 402 | 405 | 403
  Week 4, +2hr | -1.4 (8.57) | -0.3 (8.57) | -0.2 (8.01)
  Week 4, +3hr: number analyzed (Participants) | 223 | 220 | 238
  Week 4, +3hr | -0.4 (8.02) | -0.2 (8.25) | 0.2 (8.32)
  Week 4, +4hr: number analyzed (Participants) | 150 | 137 | 142
  Week 4, +4hr | 0.2 (8.79) | 0.7 (6.92) | 1.4 (8.31)
  Week 8: number analyzed (Participants) | 349 | 337 | 321
  Week 8 | 0.2 (8.15) | 0.2 (8.27) | 2.4 (8.50)
  Week 16: number analyzed (Participants) | 199 | 204 | 175
  Week 16 | -0.1 (8.06) | 0.3 (9.17) | 1.5 (9.05)
  Week 24: number analyzed (Participants) | 183 | 175 | 157
  Week 24 | 0.2 (7.91) | -0.3 (9.85) | 2.3 (8.86)
  Week 36: number analyzed (Participants) | 150 | 136 | 117
  Week 36 | 0.7 (8.27) | 0.5 (8.74) | 2.9 (8.09)
  Week 48: number analyzed (Participants) | 156 | 143 | 133
  Week 48 | 0.9 (9.01) | 1.2 (9.11) | 2.4 (8.94)
  Week 54: number analyzed (Participants) | 326 | 323 | 304
  Week 54 | -0.5 (9.33) | -0.2 (8.89) | 1.7 (8.87)

29. Secondary Outcome: Changes From Baseline in ECG Parameters- RR Interval, QT Interval, QTcB, QTcF, PR Interval and QRS Duration
Description: Triplicate 12-lead ECG measures was obtained digitally, approximately one minute apart after the participant had rested in the supine position in a quiet room (no TV, minimal talking) for atleast 10 minutes. The ECG parameters includes PR interval, QRS duration, QT - uncorrected interval, QTc Bazett (QTcB), QTc Fridericia (QTcF) and RR interval. The assessments were performed at Baseline and up to Week 54. Change from Baseline was calculated as value at scheduled time point minus Baseline value. Baseline was defined as value at Week 0. Full population data was presented.
Time Frame: Baseline (Week 0) and Weeks 4, 8, 16, 24, 36, 48, 54
Population: Safety population. Only those participants available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: MSEC
Groups:
- RSG XR 2mg: Participants randomized to this arm received Rosiglitazone 2 mg in the form of extended release (XR) once daily which remained constant throughout the 48 Week treatment period. From Week 48 all the participants received single-blind placebo treatment as one tablet daily until Visit 10 (Week 54)
Arm/Group | Placebo | RSG XR 2mg | RSG XR 8mg
Number analyzed (Participants) | 487 | 490 | 491
MSEC
  RR Interval, Week 0, +1hr: number analyzed (Participants) | 455 | 469 | 469
  RR Interval, Week 0, +1hr | 26.7 (92.91) | 17.9 (83.58) | 30.4 (92.97)
  RR Interval, Week 0, +2hr: number analyzed (Participants) | 362 | 378 | 383
  RR Interval, Week 0, +2hr | 23.8 (105.24) | 11.0 (100.67) | 17.7 (109.40)
  RR Interval, Week 0, +3hr: number analyzed (Participants) | 229 | 234 | 246
  RR Interval, Week 0, +3hr | 3.5 (103.09) | 4.6 (105.04) | 0.6 (108.88)
  RR Interval, Week 0, +4hr: number analyzed (Participants) | 163 | 145 | 155
  RR Interval, Week 0, +4hr | -8.8 (91.08) | -12.1 (92.98) | -5.7 (108.33)
  RR Interval, Week 4, Pre-Dose: number analyzed (Participants) | 443 | 442 | 443
  RR Interval, Week 4, Pre-Dose | -0.2 (99.28) | -9.6 (104.15) | -14.0 (107.71)
  RR Interval, Week 4, +1hr: number analyzed (Participants) | 429 | 435 | 437
  RR Interval, Week 4, +1hr | 23.2 (115.71) | 8.7 (115.70) | 4.3 (118.85)
  RR Interval, Week 4, +2hr: number analyzed (Participants) | 402 | 405 | 403
  RR Interval, Week 4, +2hr | 24.0 (123.53) | 6.8 (119.63) | 2.5 (122.39)
  RR Interval, Week 4, +3hr: number analyzed (Participants) | 223 | 220 | 238
  RR Interval, Week 4, +3hr | 7.4 (117.68) | 8.5 (124.69) | -3.0 (125.89)
  RR Interval, Week 4, +4hr: number analyzed (Participants) | 150 | 137 | 142
  RR Interval, Week 4, +4hr | -2.1 (117.25) | -4.7 (108.17) | -20.6 (124.14)
  RR Interval, Week 8: number analyzed (Participants) | 349 | 337 | 321
  RR Interval, Week 8 | 0.6 (110.81) | 0.5 (110.70) | -32.6 (118.98)
  RR Interval, Week 16: number analyzed (Participants) | 199 | 204 | 175
  RR Interval, Week 16 | 9.0 (110.76) | -1.5 (127.38) | -20.8 (123.59)
  RR Interval, Week 24: number analyzed (Participants) | 183 | 175 | 157
  RR Interval, Week 24 | -1.3 (119.93) | 2.8 (141.97) | -31.3 (126.48)
  RR Interval, Week 36: number analyzed (Participants) | 150 | 136 | 117
  RR Interval, Week 36 | -8.0 (114.49) | -3.7 (127.72) | -43.4 (107.83)
  RR Interval, Week 48: number analyzed (Participants) | 156 | 143 | 133
  RR Interval, Week 48 | -8.2 (125.15) | -17.0 (132.82) | -32.7 (121.98)
  RR Interval, Week 54: number analyzed (Participants) | 326 | 323 | 304
  RR Interval, Week 54 | 10.9 (128.93) | 5.4 (119.76) | -26.0 (125.53)
  QT interval, Week 0, +1hr: number analyzed (Participants) | 455 | 469 | 469
  QT interval, Week 0, +1hr | 5.2 (18.01) | 4.5 (17.29) | 5.4 (17.07)
  QT Interval, Week 0, +2hr: number analyzed (Participants) | 362 | 378 | 383
  QT Interval, Week 0, +2hr | 6.4 (19.64) | 3.8 (20.70) | 5.0 (19.62)
  QT Interval, Week 0, +3hr: number analyzed (Participants) | 229 | 234 | 246
  QT Interval, Week 0, +3hr | 2.2 (19.38) | 3.2 (20.61) | 1.9 (21.79)
  QT Interval, Week 0, +4hr: number analyzed (Participants) | 163 | 145 | 155
  QT Interval, Week 0, +4hr | -0.3 (18.65) | -1.6 (20.13) | 1.8 (20.67)
  QT Interval, Week 4, Pre-Dose: number analyzed (Participants) | 443 | 442 | 443
  QT Interval, Week 4, Pre-Dose | -0.8 (19.18) | -0.7 (20.35) | -1.7 (23.63)
  QT Interval, Week 4, +1hr: number analyzed (Participants) | 429 | 435 | 437
  QT Interval, Week 4, +1hr | 3.6 (21.53) | 2.7 (22.14) | 1.4 (23.26)
  QT Interval, Week 4, +2hr: number analyzed (Participants) | 402 | 405 | 403
  QT Interval, Week 4, +2hr | 5.2 (22.96) | 4.2 (24.09) | 3.2 (24.54)
  QT Interval, Week 4, +3hr: number analyzed (Participants) | 223 | 220 | 238
  QT Interval, Week 4, +3hr | 3.8 (22.82) | 3.6 (25.24) | 0.6 (26.70)
  QT Interval, Week 4, +4hr: number analyzed (Participants) | 150 | 137 | 142
  QT Interval, Week 4, +4hr | 1.9 (25.13) | 0.8 (22.66) | -1.4 (25.73)
  QT Interval, Week 8: number analyzed (Participants) | 349 | 337 | 321
  QT Interval, Week 8 | -1.4 (21.30) | 0.5 (21.60) | -4.1 (24.46)
  QT Interval, Week 16: number analyzed (Participants) | 199 | 204 | 175
  QT Interval, Week 16 | 2.4 (23.39) | -0.3 (24.52) | -1.3 (25.71)
  QT Interval, Week 24: number analyzed (Participants) | 183 | 175 | 157
  QT Interval, Week 24 | 1.6 (24.35) | 2.4 (25.99) | -2.2 (25.06)
  QT Interval, Week 36: number analyzed (Participants) | 150 | 136 | 117
  QT Interval, Week 36 | 0.5 (21.85) | 0.0 (23.58) | -4.7 (27.25)
  QT Interval, Week 48: number analyzed (Participants) | 156 | 143 | 133
  QT Interval, Week 48 | 2.0 (24.53) | -0.7 (26.19) | -2.7 (29.56)
  QT Interval, Week 54: number analyzed (Participants) | 326 | 323 | 304
  QT Interval, Week 54 | 2.1 (24.97) | 2.4 (23.41) | -1.2 (25.41)
  QTcB interval, Week 0, +1hr: number analyzed (Participants) | 155 | 469 | 469
  QTcB interval, Week 0, +1hr | -0.4 (13.49) | 0.7 (14.41) | -0.7 (14.02)
  QTcB Interval, Week 0, +2hr: number analyzed (Participants) | 362 | 378 | 383
  QTcB Interval, Week 0, +2hr | 1.6 (14.35) | 1.6 (15.70) | 1.5 (15.68)
  QTcB Interval, Week 0, +3hr: number analyzed (Participants) | 229 | 234 | 246
  QTcB Interval, Week 0, +3hr | 1.9 (15.19) | 2.4 (15.73) | 2.0 (14.60)
  QTcB Interval, Week 0, +4hr: number analyzed (Participants) | 163 | 145 | 155
  QTcB Interval, Week 0, +4hr | 1.7 (13.48) | 1.2 (19.50) | 3.2 (14.99)
  QTcB Interval, Week 4, Pre-Dose: number analyzed (Participants) | 443 | 442 | 443
  QTcB Interval, Week 4, Pre-Dose | -0.5 (15.98) | 1.3 (17.14) | 1.5 (18.50)
  QTcB Interval, Week 4, +1hr: number analyzed (Participants) | 429 | 435 | 437
  QTcB Interval, Week 4, +1hr | -0.9 (16.84) | 0.9 (17.51) | 1.0 (16.88)
  QTcB Interval, Week 4, +2hr: number analyzed (Participants) | 402 | 405 | 403
  QTcB Interval, Week 4, +2hr | 0.4 (17.13) | 2.8 (16.73) | 2.9 (17.74)
  QTcB Interval, Week 4, +3hr: number analyzed (Participants) | 223 | 220 | 238
  QTcB Interval, Week 4, +3hr | 2.4 (18.56) | 2.1 (17.72) | 1.6 (17.87)
  QTcB Interval, Week 4, +4hr: number analyzed (Participants) | 150 | 137 | 142
  QTcB Interval, Week 4, +4hr | 2.8 (17.83) | 2.3 (20.30) | 3.6 (15.95)
  QTcB Interval, Week 8: number analyzed (Participants) | 349 | 337 | 321
  QTcB Interval, Week 8 | -1.3 (15.27) | 0.7 (18.78) | 3.2 (18.09)
  QTcB Interval, Week 16: number analyzed (Participants) | 199 | 204 | 175
  QTcB Interval, Week 16 | 1.1 (18.12) | 0.3 (18.73) | 3.6 (16.81)
  QTcB Interval, Week 24: number analyzed (Participants) | 183 | 175 | 157
  QTcB Interval, Week 24 | 2.2 (19.04) | 1.5 (18.81) | 5.2 (17.97)
  QTcB Interval, Week 36: number analyzed (Participants) | 150 | 136 | 117
  QTcB Interval, Week 36 | 2.5 (17.87) | 0.9 (19.37) | 4.3 (19.16)
  QTcB Interval, Week 48: number analyzed (Participants) | 156 | 143 | 133
  QTcB Interval, Week 48 | 4.5 (18.91) | 3.1 (18.34) | 5.0 (18.39)
  QTcB Interval, Week 54: number analyzed (Participants) | 326 | 323 | 304
  QTcB Interval, Week 54 | 0.2 (18.42) | 1.4 (18.74) | 4.5 (18.67)
  QTcF interval, Week 0, +1hr: number analyzed (Participants) | 455 | 469 | 469
  QTcF interval, Week 0, +1hr | 1.5 (11.92) | 2.0 (12.78) | 1.3 (11.99)
  QTcF Interval, Week 0, +2hr: number analyzed (Participants) | 362 | 378 | 383
  QTcF Interval, Week 0, +2hr | 3.2 (12.50) | 2.3 (14.24) | 2.6 (13.08)
  QTcF Interval, Week 0, +3hr: number analyzed (Participants) | 229 | 234 | 246
  QTcF Interval, Week 0, +3hr | 1.9 (13.34) | 2.6 (13.89) | 1.9 (13.44)
  QTcF Interval, Week 0, +4hr: number analyzed (Participants) | 163 | 145 | 155
  QTcF Interval, Week 0, +4hr | 1.0 (12.31) | 0.2 (17.24) | 2.8 (12.93)
  QTcF Interval, Week 4, Pre-Dose: number analyzed (Participants) | 443 | 442 | 443
  QTcF Interval, Week 4, Pre-Dose | -0.6 (13.82) | 0.6 (14.80) | 0.4 (17.02)
  QTcF Interval, Week 4, +1hr: number analyzed (Participants) | 429 | 435 | 437
  QTcF Interval, Week 4, +1hr | 0.6 (14.45) | 1.5 (15.13) | 1.1 (15.15)
  QTcF Interval, Week 4, +2hr: number analyzed (Participants) | 402 | 405 | 403
  QTcF Interval, Week 4, +2hr | 2.0 (14.65) | 3.3 (15.10) | 2.9 (16.01)
  QTcF Interval, Week 4, +3hr: number analyzed (Participants) | 223 | 220 | 238
  QTcF Interval, Week 4, +3hr | 2.9 (16.15) | 2.6 (16.19) | 1.3 (16.97)
  QTcF Interval, Week 4, +4hr: number analyzed (Participants) | 150 | 137 | 142
  QTcF Interval, Week 4, +4hr | 2.5 (16.51) | 1.7 (17.88) | 1.9 (15.19)
  QTcF Interval, Week 8: number analyzed (Participants) | 349 | 337 | 321
  QTcF Interval, Week 8 | -1.4 (13.29) | 0.6 (15.94) | 0.7 (16.39)
  QTcF Interval, Week 16: number analyzed (Participants) | 199 | 204 | 175
  QTcF Interval, Week 16 | 1.4 (16.62) | 0.1 (16.20) | 1.9 (15.77)
  QTcF Interval, Week 24: number analyzed (Participants) | 183 | 175 | 157
  QTcF Interval, Week 24 | 2.0 (17.21) | 1.9 (16.00) | 2.6 (15.84)
  QTcF Interval, Week 36: number analyzed (Participants) | 150 | 136 | 117
  QTcF Interval, Week 36 | 1.8 (15.23) | 0.6 (16.22) | 1.3 (19.30)
  QTcF Interval, Week 48: number analyzed (Participants) | 156 | 143 | 133
  QTcF Interval, Week 48 | 3.5 (16.61) | 1.8 (16.49) | 2.4 (18.86)
  QTcF Interval, Week 54: number analyzed (Participants) | 326 | 323 | 304
  QTcF Interval, Week 54 | 0.8 (16.08) | 1.7 (15.93) | 2.6 (16.74)
  PR Interval, Week 0, +1hr: number analyzed (Participants) | 437 | 449 | 450
  PR Interval, Week 0, +1hr | 0.6 (10.45) | 0.0 (10.39) | 0.4 (10.00)
  PR Interval, Week 0, +2hr: number analyzed (Participants) | 349 | 364 | 366
  PR Interval, Week 0, +2hr | 0.0 (10.82) | 0.2 (11.79) | -0.8 (10.97)
  PR Interval, Week 0, +3hr: number analyzed (Participants) | 220 | 226 | 234
  PR Interval, Week 0, +3hr | 0.2 (10.74) | -0.1 (11.02) | -0.8 (11.78)
  PR Interval, Week 0, +4hr: number analyzed (Participants) | 155 | 136 | 149
  PR Interval, Week 0, +4hr | 1.8 (12.62) | 1.5 (10.47) | 0.0 (11.04)
  PR Interval, Week 1, Pre-dose: number analyzed (Participants) | 427 | 420 | 424
  PR Interval, Week 1, Pre-dose | -0.2 (12.81) | 0.4 (13.78) | 0.7 (11.51)
  PR Interval, Week 1, +1hr: number analyzed (Participants) | 415 | 412 | 418
  PR Interval, Week 1, +1hr | 0.3 (13.50) | 1.6 (13.43) | 1.3 (11.73)
  PR Interval, Week 1, +2hr: number analyzed (Participants) | 389 | 386 | 385
  PR Interval, Week 1, +2hr | 0.7 (13.27) | 0.9 (12.17) | 1.5 (11.98)
  PR Interval, Week 1, +3hr: number analyzed (Participants) | 216 | 211 | 228
  PR Interval, Week 1, +3hr | 0.7 (14.43) | 1.4 (13.81) | 2.6 (12.96)
  PR Interval, Week 1, +4hr: number analyzed (Participants) | 145 | 130 | 138
  PR Interval, Week 1, +4hr | 0.9 (15.31) | 1.1 (15.56) | 0.8 (11.62)
  PR Interval, Week 8: number analyzed (Participants) | 338 | 319 | 310
  PR Interval, Week 8 | -1.3 (13.20) | 0.7 (11.94) | 0.8 (12.52)
  PR Interval, Week 16: number analyzed (Participants) | 193 | 191 | 167
  PR Interval, Week 16 | -0.7 (15.22) | 0.6 (12.00) | 0.1 (15.06)
  PR Interval, Week 24: number analyzed (Participants) | 178 | 166 | 152
  PR Interval, Week 24 | -1.9 (12.43) | 0.1 (12.28) | -0.5 (13.38)
  PR Interval, Week 36: number analyzed (Participants) | 142 | 128 | 114
  PR Interval, Week 36 | -1.2 (13.87) | -2.3 (12.25) | -0.9 (13.70)
  PR Interval, Week 48: number analyzed (Participants) | 148 | 136 | 130
  PR Interval, Week 48 | -0.6 (16.83) | -2.5 (13.48) | -0.8 (12.99)
  PR Interval, Week 54: number analyzed (Participants) | 313 | 307 | 294
  PR Interval, Week 54 | -0.5 (13.66) | -0.6 (13.47) | 0.0 (11.99)
  QRS Interval, Week 0, +1hr: number analyzed (Participants) | 455 | 469 | 469
  QRS Interval, Week 0, +1hr | 0.2 (5.49) | 0.6 (6.26) | 0.4 (5.64)
  QRS Interval, Week 0, +2hr: number analyzed (Participants) | 362 | 378 | 383
  QRS Interval, Week 0, +2hr | 0.2 (5.44) | 0.8 (6.82) | 0.4 (5.61)
  QRS Interval, Week 0, +3hr: number analyzed (Participants) | 229 | 234 | 246
  QRS Interval, Week 0, +3hr | -0.1 (5.30) | 0.8 (6.34) | 0.5 (6.20)
  QRS Interval, Week 0, +4hr: number analyzed (Participants) | 163 | 145 | 155
  QRS Interval, Week 0, +4hr | 0.1 (5.72) | 0.5 (7.95) | -0.2 (6.15)
  QRS Interval, Week 4, Pre-Dose: number analyzed (Participants) | 443 | 442 | 443
  QRS Interval, Week 4, Pre-Dose | 0.6 (7.45) | 0.2 (7.91) | 0.8 (7.38)
  QRS Interval, Week 4, +1hr: number analyzed (Participants) | 429 | 435 | 437
  QRS Interval, Week 4, +1hr | 1.1 (7.17) | 0.4 (8.44) | 1.0 (7.51)
  QRS Interval, Week 4, +2hr: number analyzed (Participants) | 402 | 405 | 403
  QRS Interval, Week 4, +2hr | 1.0 (7.60) | 0.7 (7.87) | 1.5 (7.71)
  QRS Interval, Week 4, +3hr: number analyzed (Participants) | 223 | 220 | 238
  QRS Interval, Week 4, +3hr | 1.3 (8.86) | 0.7 (7.48) | 1.5 (8.08)
  QRS Interval, Week 4, +4hr: number analyzed (Participants) | 150 | 137 | 142
  QRS Interval, Week 4, +4hr | 0.1 (9.19) | 0.8 (9.10) | 1.4 (9.12)
  QRS Interval, Week 8: number analyzed (Participants) | 349 | 337 | 321
  QRS Interval, Week 8 | 0.2 (7.17) | 0.8 (7.15) | 0.5 (8.26)
  QRS Interval, Week 16: number analyzed (Participants) | 199 | 204 | 175
  QRS Interval, Week 16 | 0.8 (8.91) | -0.5 (8.42) | 0.1 (6.96)
  QRS Interval, Week 24: number analyzed (Participants) | 183 | 175 | 157
  QRS Interval, Week 24 | 0.9 (8.72) | 1.3 (8.02) | 1.1 (6.71)
  QRS Interval, Week 36: number analyzed (Participants) | 150 | 136 | 117
  QRS Interval, Week 36 | 1.7 (9.14) | 1.7 (12.81) | 0.4 (6.66)
  QRS Interval, Week 48: number analyzed (Participants) | 156 | 143 | 133
  QRS Interval, Week 48 | 1.5 (9.52) | 1.3 (11.52) | 1.0 (7.19)
  QRS Interval, Week 54: number analyzed (Participants) | 326 | 323 | 304
  QRS Interval, Week 54 | 0.8 (9.29) | 0.9 (9.40) | 1.1 (8.28)

30. Secondary Outcome: Change From Baseline in HbA1c up to Week 54
Description: Blood samples were collected for assessments of HbA1c levels at Baseline, Weeks 12, 24, 36, 48, 54. Change from Baseline was calculated as value at scheduled time point minus Baseline value. Baseline was defined as value at Week 0.
Time Frame: Baseline (Week 0) and Weeks 12, 24, 36, 48, 54
Population: Safety population. Only those participants available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Percentage of HbA1c
Arm/Group | Placebo | RSG XR 2mg | RSG XR 8mg
Number analyzed (Participants) | 487 | 490 | 491
Percentage of HbA1c
  Week 12: number analyzed (Participants) | 107 | 86 | 79
  Week 12 | 0.02 (0.300) | 0.13 (0.278) | 0.15 (0.398)
  Week 24: number analyzed (Participants) | 152 | 147 | 133
  Week 24 | 0.09 (0.370) | 0.17 (0.415) | 0.17 (0.422)
  Week 36: number analyzed (Participants) | 125 | 127 | 107
  Week 36 | 0.15 (0.398) | 0.19 (0.273) | 0.25 (0.418)
  Week 48: number analyzed (Participants) | 339 | 326 | 309
  Week 48 | 0.16 (0.394) | 0.19 (0.323) | 0.27 (0.400)
  Week 54: number analyzed (Participants) | 19 | 20 | 22
  Week 54 | 0.09 (0.346) | 0.03 (0.483) | 0.03 (0.338)

31. Secondary Outcome: Change From Baseline in Short Term Memory Assessment
Description: The 11-item ADAS-Cog assessed a range of cognitive abilities including memory, comprehension, orientation in time and place and spontaneous speech. Most items were evaluated by tests, but some were dependent on clinician ratings on a five point scale. Scores range from 0 to 70 with higher scores indicating greater dysfunction. Questions 1 (word recall) and 7 (word recognition) of ADAS-Cog questionnaire was summed to get a short term memory assessment. The score for Question 1 was calculated as the mean number of words not recalled over the trials for which data was available. If data for all three trials was missing, or if the score for Question 7 was missing then the short term memory score will also be set to missing. Change from Baseline was calculated as value at scheduled time point minus Baseline value. Baseline was defined as value a t Week 0. Estimated value was calculated by Active treatment minus Placebo. The adjusted means were presented.
Time Frame: Baseline (Week 0) and upto Week 48
Population: ITT population. Number of participants with observed data contributing to the analysis.
Measure: Least Squares Mean (Standard Error); unit: Scores on an scale
Arm/Group | Placebo | RSG XR 2mg | RSG XR 8mg
Number analyzed (Participants) | 479 | 480 | 470
Scores on an scale
  Week 8: number analyzed (Participants) | 453 | 449 | 437
  Week 8 | -0.2 (0.14) | -0.2 (0.14) | -0.1 (0.13)
  Week 16: number analyzed (Participants) | 433 | 423 | 406
  Week 16 | -0.3 (0.14) | -0.4 (0.14) | -0.5 (0.13)
  Week 24: number analyzed (Participants) | 414 | 401 | 373
  Week 24 | -0.0 (0.15) | -0.0 (0.15) | 0.2 (0.14)
  Week 36: number analyzed (Participants) | 376 | 374 | 349
  Week 36 | 0.6 (0.15) | 0.7 (0.15) | 0.7 (0.15)
  Week 48: number analyzed (Participants) | 354 | 335 | 329
  Week 48 | 0.6 (0.16) | 0.6 (0.17) | 0.9 (0.16)
Statistical Analysis 1: Comparison: Placebo vs RSG XR 2mg; For Week 8; Test type: Superiority; p = 0.748, Mixed model for repeated measures; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Net) = -0.1, 95% CI 2-sided [-0.4 to 0.3] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs RSG XR 8mg; For Week 8; Test type: Superiority; p = 0.617, Mixed model for repeated measures; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Net) = 0.1, 95% CI 2-sided [-0.3 to 0.5] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs RSG XR 2mg; Week 16; Test type: Superiority; p = 0.708, Mixed model for repeated measures; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Net) = -0.1, 95% CI 2-sided [-0.5 to 0.3] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Placebo vs RSG XR 8mg; Week 16; Test type: Superiority; p = 0.400, Mixed model for repeated measures; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Net) = -0.2, 95% CI 2-sided [-0.5 to 0.2] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Placebo vs RSG XR 2mg; For Week 24; Test type: Superiority; p = 0.928, Mixed model for repeated measures; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Net) = 0.0, 95% CI 2-sided [-0.4 to 0.4] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Placebo vs RSG XR 8mg; For Week 24; Test type: Superiority; p = 0.178, Mixed model for repeated measures; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Net) = 0.3, 95% CI 2-sided [-0.1 to 0.7] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: Placebo vs RSG XR 2mg; For Week 36; Test type: Superiority; p = 0.626, Mixed model for repeated measures; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Net) = 0.1, 95% CI 2-sided [-0.3 to 0.5] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 8: Comparison: Placebo vs RSG XR 8mg; For Week 36; Test type: Superiority; p = 0.608, Mixed model for repeated measures; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Net) = 0.1, 95% CI 2-sided [-0.3 to 0.5] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 9: Comparison: Placebo vs RSG XR 2mg; For Week 48; Test type: Superiority; p = 0.865, Mixed model for repeated measures; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Net) = 0.0, 95% CI 2-sided [-0.5 to 0.4] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 10: Comparison: Placebo vs RSG XR 8mg; For Week 48; Test type: Superiority; p = 0.149, Mixed model for repeated measures; Mixed model for repeated measures with restricted maximum likelihood estimation and an unstructured covariance matrix; Mean Difference (Net) = 0.3, 95% CI 2-sided [-0.1 to 0.8] — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-serious AEs were collected from the first dose of investigational product until Week 54 following early withdrawal of the study medication/follow up
Description: Serious adverse events (SAEs) and non-serious AEs were collected safety population (full population cohort), comprised of all randomized participants who received at least one dose of study medication.
Arm/Group | Placebo | RSG XR 2mg | RSG XR 8mg
All-Cause Mortality (participants affected / at risk) | 9/487 | 11/490 | 11/491
Serious Adverse Events (participants affected / at risk) | 60/487 | 58/490 | 66/491
Other Adverse Events (participants affected / at risk) | 11/487 | 42/490 | 100/491
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=487) | RSG XR 2mg (N=490) | RSG XR 8mg (N=491)
Syncope (Nervous system disorders) | 5 | 1 | 3
Cerebrovascular accident (Nervous system disorders) | 1 | 3 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 1 | 1
Convulsion (Nervous system disorders) | 1 | 0 | 1
Loss of consciousness (Nervous system disorders) | 0 | 1 | 1
Nervous system disorder (Nervous system disorders) | 0 | 2 | 0
Cerebral haematoma (Nervous system disorders) | 1 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 1 | 0
Cerebral hypoperfusion (Nervous system disorders) | 0 | 0 | 1
Cerebral infarction (Nervous system disorders) | 1 | 0 | 0
Cerebral ischaemia (Nervous system disorders) | 0 | 1 | 0
Dementia Alzheimer's type (Nervous system disorders) | 0 | 0 | 1
Depressed level of consciousness (Nervous system disorders) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 0
Encephalopathy (Nervous system disorders) | 0 | 1 | 0
Epilepsy (Nervous system disorders) | 0 | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 1
Metabolic encephalopathy (Nervous system disorders) | 1 | 0 | 0
Reversible ischaemic neurological deficit (Nervous system disorders) | 0 | 0 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 0 | 0
Syncope vasovagal (Nervous system disorders) | 0 | 1 | 0
Tonic convulsion (Nervous system disorders) | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 3 | 3 | 1
Hip fracture (Injury, poisoning and procedural complications) | 3 | 1 | 2
Femur fracture (Injury, poisoning and procedural complications) | 2 | 0 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 2 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Carbon monoxide poisoning (Injury, poisoning and procedural complications) | 1 | 0 | 0
Cardiac pacemaker malfunction (Injury, poisoning and procedural complications) | 1 | 0 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Exposure to toxic agent (Injury, poisoning and procedural complications) | 0 | 1 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Forearm fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Fractured ischium (Injury, poisoning and procedural complications) | 0 | 1 | 0
Ilium fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Post procedural pulmonary embolism (Injury, poisoning and procedural complications) | 0 | 1 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0
Soft tissue injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 3 | 3
Bronchitis (Infections and infestations) | 2 | 1 | 3
Urinary tract infection (Infections and infestations) | 0 | 1 | 3
Cystitis (Infections and infestations) | 1 | 0 | 1
Bronchopneumonia (Infections and infestations) | 1 | 0 | 0
Bursitis infective (Infections and infestations) | 0 | 0 | 1
Encephalitis herpes (Infections and infestations) | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Meningitis viral (Infections and infestations) | 0 | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 1 | 0
Pyelonephritis acute (Infections and infestations) | 1 | 0 | 0
Pyelonephritis chronic (Infections and infestations) | 0 | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0
Septic shock (Infections and infestations) | 0 | 1 | 0
Urosepsis (Infections and infestations) | 0 | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 0 | 3
Myocardial infarction (Cardiac disorders) | 1 | 0 | 3
Arrhythmia (Cardiac disorders) | 0 | 2 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 1
Atrioventricular block (Cardiac disorders) | 1 | 0 | 0
Atrioventricular block complete (Cardiac disorders) | 0 | 1 | 0
Bradycardia (Cardiac disorders) | 0 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 1 | 0
Left ventricular failure (Cardiac disorders) | 0 | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 0 | 1 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 1
Right ventricular failure (Cardiac disorders) | 0 | 0 | 1
Sick sinus syndrome (Cardiac disorders) | 1 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 0 | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Lip neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Salivary gland cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 2 | 1 | 0
Abnormal behaviour (Psychiatric disorders) | 0 | 1 | 1
Hallucination (Psychiatric disorders) | 1 | 1 | 0
Adjustment disorder (Psychiatric disorders) | 0 | 0 | 1
Aggression (Psychiatric disorders) | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0
Bipolar disorder (Psychiatric disorders) | 1 | 0 | 0
Mental disorder due to a general medical condition (Psychiatric disorders) | 0 | 0 | 1
Psychotic disorder (Psychiatric disorders) | 1 | 0 | 0
Melaena (Gastrointestinal disorders) | 0 | 1 | 1
Abdominal hernia (Gastrointestinal disorders) | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0
Food poisoning (Gastrointestinal disorders) | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1
Lip oedema (Gastrointestinal disorders) | 0 | 1 | 0
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Bronchopneumopathy (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Death (General disorders) | 0 | 0 | 1
General physical health deterioration (General disorders) | 0 | 0 | 1
Generalised oedema (General disorders) | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 0 | 1
Sudden cardiac death (General disorders) | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 2
Orthostatic hypotension (Vascular disorders) | 0 | 1 | 1
Aortic aneurysm (Vascular disorders) | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0
Bile duct stenosis (Hepatobiliary disorders) | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0
Cholestasis (Hepatobiliary disorders) | 1 | 0 | 0
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 0 | 1
Renal colic (Renal and urinary disorders) | 1 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 1 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 1
Cataract (Eye disorders) | 1 | 0 | 0
Weight decreased (Investigations) | 1 | 0 | 0
Epididymitis (Reproductive system and breast disorders) | 1 | 0 | 0
Lordosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=487) | RSG XR 2mg (N=490) | RSG XR 8mg (N=491)
Oedema peripheral (General disorders) | 9 | 32 | 91
Anaemia (Blood and lymphatic system disorders) | 2 | 10 | 25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.